Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

**CC Protocol #:** 16-C-0048

OSP#: 1511-1478

**NCT** #: NCT02649855

IBC#: RD-15-IX-08 Version Date: August 8, 2018

Amendment: H

Title: Docetaxel and PROSTVAC for Metastatic Castration Sensitive Prostate Cancer

Ravi Madan, M.D. NCI Principal Investigator:

Genitourinary Malignancies Branch (GMB), CCR, NCI

Building 10, Rm. 13N240

Bethesda, MD 20892

Phone: 301-480-7168

Email: madanr@mail.nih.gov

Epic Sciences F, G Collaborator:

Attn: Ryan Dittamore

9381 Judicial Drive, Suite 200

San Diego, CA 92121

Phone: 858-356-6610, ext. 124

Email: ryan.dittamore@epicsciences.com

#### Investigational Agents:

| Drug Name | PROSTVAC-V/F |
|------------|---------------------------------|
| IND Number | 15455 |
| Sponsor | Center for Cancer Research, NCI |

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

| Manufacturer | Bavarian Nordic, Inc. |
|--------------|-----------------------|
| Supplier | Bavarian Nordic, Inc. |

#### Commercial Agents:

Docetaxel will be obtained from commercial sources by the local site pharmacy.

#### **PRÉCIS**

#### Background:

- survival (57.6 vs 44.0 months (HR=0.56, (0.44-0.70), p <0.0001) for men with metastatic castration sensitive prostate cancer A phase III trial demonstrated that combining docetaxel and androgen deprivation therapy (ADT) significantly improved
- PROSTVAC (developed by the National Cancer Institute [NCI] and licensed to Bavarian Nordic Immunotherapeutics, Mountain View, CA) is a therapeutic cancer vaccine for prostate cancer.
- Preclinical and clinical studies support the potential synergy in the combination of docetaxel and PROSTVAC. The potential to combine docetaxel with vaccine in mCSPC could improve upon the survival advantage that has been previously seen.

#### Objectives:

Primary

To determine if PROSTVAC combined with docetaxel is able to induce greater antigen spreading (i.e. a broader immune response) with greater associated response score compared to docetaxel alone after 19 weeks.

#### Key Eligibility Criteria:

- Must have castrate sensitive prostate cancer (rising PSA and testosterone over 100) or is within 134 days of starting ADT (Arm A or B) or within 28 days of start ADT (Arm C)
- Histopathological confirmation of prostate cancer
- Patients must have metastatic disease
- Patients must have a performance status of 0 to 2 according to the ECOG criteria
- Patients must have adequate bone marrow, hepatic, and renal function

#### Design

- weeks x 6 cycles versus ADT followed by sequential docetaxel 75 mg/m2 q3 weeks x 6 cycles followed by PROSTVAC q3 This is a randomized trial of ADT followed by simultaneous docetaxel 75 mg/m2 q3 weeks x 6 cycles + PROSTVAC q3 weeks x 6 cycles in men with newly diagnosed mCSPC.
- Patients who have not started ADT or who have been on ADT 28 days or fewer will be assigned to treatment with PROSTVAC for 4 -6 injections followed by docetaxel 75 mg/m2 q3 weeks x 6 cycles.

#### SCHEMA

#### Arm A and Arm B

Version Date: 8/8/18 Abbreviated Title: Docetaxel & PROSTVAC in mCSPC



#### Arm C

for 6 injections followed by docetaxel 75 mg/m2 q3 weeks x 6 cycles. Investigator may use clinical discretion to start docetaxel after Patients who have not started ADT or who have been on ADT for less than 28 days will be assigned to treatment with PROSTVAC 4 vaccines (e.g. 1 dose of vaccinia-PROSTVAC, followed by 3 doses of fowlpox-PROSTVAC).

#### Version Date: 8/8/18 Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

#### TABLE OF CONTENTS

| PRÉCIS | | 7 |
|---|---|---|
| SCHE | SCHEMA | |
| TABL | TABLE OF CONTENTS | · · · |
| 1 IP | INTRODUCTION | 7 |
| 1.1 | Study Objectives | 7 |
| 1.2 | Background and Rationale | ∞<br>: |
| 2 E | ELIGIBILITY ASSESSMENT AND ENROLLMENT | . 23 |
| 2.1 | Eligibility Criteria | . 23 |
| 2.2 | Screening Evaluation. | . 26 |
| 2.3 | Baseline Evaluation | . 27 |
| 2.4 | Registration Procedures | . 28 |
| 3 S | STUDY IMPLEMENTATION | . 30 |
| 3.1 | Study Design . | . 30 |
| 3.2 | Drug Administration | . 30 |
| 3.3 | Criteria for Removal from Protocol Therapy and Off Study Criteria | . 34 |
| 3.4 | Follow-up Evaluations | . 35 |
| 3.5 | Post-Study Evaluation | . 36 |
| 4<br>O | CONCOMITANT MEDICATIONS/MEASURES | . 36 |
| 4.1 | Concurrent Medications/Interventions | .37 |
| 4.2 | Treatment of Vaccinia Vaccination Complications | . 38 |
| 5 Bj | Biospecimen collection | . 39 |

## Version Date: 8/8/18 Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

| 2 | 5.1 C | Correlative studies for research/pharmacokinetic studies | 36 |
|---|---|---|---|
| 5 | 5.2 B | Biomarker Studies | 4 |
| 5 | 5.3 S | Sample Storage, Tracking and Disposition | 4, |
| | DAT | | 4 |
| 9 | 6.1 L | Data Collection. | 4 |
| 9 | 6.2 D | Data Sharing Plans | 2( |
| 9 | 6.3 R | Response Criteria | 2( |
| 9 | 6.4 T | Toxicity Criteria | 5 |
| 9 | 6.5 A | Antigen Spread Scoring | 5 |
| _ | SAFI | SAFETY REPORTING REQUIREMENTS/DATA AND SAFETY MONITORING PLAN | 9 |
| 7 | 7.1 D | Definitions | )9 |
| 7 | .2 N | NIH-IRB and Clinical Director (CD) Reporting | 9 |
| 7 | 7.3 II | IND Sponsor Reporting Criteria | 9 |
| 7 | 7.4 S | Safety Reporting Criteria to the Pharmaceutical Collaborators | 9 |
| 7 | 7.5 I <sub>1</sub> | Institutional Biosafety Committee (IBC) Reporting Criteria | 9 |
| 7 | 7.6 L | Data and Safety Monitoring Plan | 99 |
| 20 | STA | STATISTICAL CONSIDERATIONS | 9 |
| <b>∞</b> | 8.1 A | Arms A and B | 9 |
| <b>∞</b> | 8.2 A | Arm C. | 39 |
| <b>∞</b> | 8.3 A | Accrual | 59 |
| | COL | COLLABORATIVE AGREEMENTS | 59 |
| 6 | 9.1 A | Agreement Type | 59 |
| 0 | HUM | 0 HUMAN SUBJECTS PROTECTIONS | $\sim$ |

| 10.1 | Kationale For Subject Selection | |
|---|---|---|
| 10.3 | Participation of Children | 7 |
| 10.4 | Participation of Subjects Unable to Give Consent | 7 |
| 10.5 | Evaluation of Benefits and Risks/Discomforts | 7 |
| 10.6 | Risks/Benefits Analysis | 72 |
| 10.7 | Consent and Assent Process and Documentation | 7 |
| 1 PF | PHARMACEUTICAL INFORMATION. | 73 |
| 11.1 | Recombinant Fowlpox-PSA(L155)TRICOM <sup>TM</sup> | 73 |
| 11.2 | Recombinant Vaccinia-PSA(L155)/TRICOM <sup>TM</sup> | 7 |
| 11.3 | Docetaxel (TAXOTERE®) | <b>∞</b> |
| 2 RI | REFERENCES | 9 |
| 3 A <sub>I</sub> | Appendix A: Study Calendar | 6: |
| 4 A <sub>I</sub> | Appendix B: Performance Status Criteria | 100 |
| 5 A <sub>I</sub> | Appendix C: Vaccinia-PROSTVAC Patient Instruction Sheet | 10 |
| 6 Ag | Appendix D: Guidelines for Prophylaxis and Treatment for Hypersensitivity Reactions (HSR) Associated with Docetaxel | 107 |

#### INTRODUCTION

#### 1.1 STUDY OBJECTIVES

#### 1.1.1 Primary Objectives:

• To determine if PROSTVAC combined with docetaxel is able to induce greater antigen spreading (i.e. a broader immune response) with greater associated response score as defined in section 1.2.5 compared to docetaxel alone after 19 weeks.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

### 1.1.2 Secondary Objectives:

- Evaluate immunologic response among immune subsets (flow cytometry).
- Evaluate antigen-specific immune responses and response scores at 39 weeks in both groups and 1 year in both groups.
- Compare antigen-specific immune responses and response scores at 19 weeks in the combination arm (docetaxel and PROSTVAC) and compared to 39 weeks in the sequence arm (docetaxel followed by PROSTVAC)
- In addition, patients getting PROSTVAC prior to chemotherapy will be evaluated for antigen specific responses after completing vaccine followed by 6 cycles of chemotherapy.
- Evaluate radiographic and biochemical time to progression in all groups.
- Evaluate proportion of patients with PSA >0.2 ng/ml at 6 and 12 months.
- Evaluate changes in the tumor microenvironment with biopsies pre and post (2 cycles of vaccine therapy; alone or combination) when feasible (Biopsies could include primary tumor.)
- Evaluate pharmacogenomic studies to evaluate drug metabolism and transporters.
- Evaluate overall survival.
- The scores from the subset consisting of previously untreated patients on the superior randomized arm will be tested against the patients on the new PROSTVAC then docetaxel arm (Arm C).

## 1.2 BACKGROUND AND RATIONALE

Among the approximately 220,000 men diagnosed each year with prostate cancer in the United States, approximately 10% of them will be diagnosed with metastatic disease. [1] In addition, for the approximately 90,000 men who cannot be cured of their prostate cancer, many of them will also develop metastatic disease before the initiation of androgen deprivation therapy (ADT).  $[\underline{2}]$  Until recently, ADT was the only standard of care for patients with metastatic castration prostate cancer (mCSPC) ECOG 3805 was designed to evaluate docetaxel (for six 3-week cycles) with ADT in patients with mCSPC. (Patients were allowed to 0.70), p <0.0001). [3] Recently, a second similar study has supported these findings demonstrating an improvement in survival when 57.6 vs. 44.0 months (HR=0.61 (0.47-0.80), p=0.0003). In addition, patients treated with ADT+docetaxel for six 3-week cycles there have started ADT within 120 days of starting Docetaxel.) The results of the study indicated that docetaxel extended overall survival a comparable population of patients received six cycles of docetaxel plus standard of care compared to standard of care alone (65 vs. was a delay in progression (development of metastatic castration resistant prostate cancer) of 20.7 vs. 14.7 months (HR=0.56, (0.44-

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

43 months; HR=0.73(0.59-0.89), p=0.002). [4] Based on the findings of this study, six cycles of docetaxel + ADT is now a standard of care for patients with mCSPC

(generated from preclinical and clinical studies done here at the NCI within GMB and LTIB) that the benefits of docetaxel could be With this new available standard of care option, there is interest to build on these findings. Furthermore, there is a strong rationale enhanced by immunotherapy combinations.

## 1.2.1 Immunotherapy in Prostate Cancer

Sipuleucel-T is a therapeutic cancer vaccine generated from peripheral blood mononuclear cells obtained from individual patients via regional processing center where they are exposed in vitro to a PAP/GM-CSF fusion protein. At the end of this process, the activated phase III trial (n = 512) demonstrated an overall survival benefit for the vaccine (25.8 months vs. 21.7 months; P = 0.032). [ $\overline{6}$ ] Based cellular product is re-infused into the patient. A full course of therapy repeats this process 3 times every 2 weeks for 1 month. [5] A The goal of therapeutic cancer vaccines is to generate a targeted immune response leading to immune-mediated anti-tumor activity. leukapheresis. This vaccine is generated after a patient's peripheral immune cells are collected via leukapheresis, transported to a on these overall survival findings, the FDA approved sipuleucel-T for the treatment of asymptomatic or minimally symptomatic mCRPC, making it the first FDA-approved therapeutic cancer vaccine for the treatment of any malignancy

#### PROSTVAC

(PSA), PROSTVAC vaccine employs genetically altered poxviruses to generate an immune response. Administered subcutaneously, expressing a PSA peptide within the major histocompatibility complex, resulting in PSA-specific cytolytic T lymphocytes activation. PROSTVAC (PROSTVAC<sup>TM</sup>; developed by the National Cancer Institute [NCI] and licensed to Bavarian Nordic, Mountain View, Nordic have an ongoing CRADA for the preclinical and clinical development of PROSTVAC.) To target prostate-specific antigen the poxviruses deliver the transgenes for the tumor associated antigens (PSA) to antigen presenting cells through cellular infection. Once these pox viruses are within the cellular cytoplasm, the transgenes are processed. The end result is an antigen presenting cell CA), an off-the-shelf therapeutic cancer vaccine, offers an alternative strategy to sipuleucel-T. [2, 8] (The LTIB and Bavarian [8] (Figure 1) This approach does not require expensive, labor-intensive ex vivo preparation of patients' peripheral blood PROSTVAC is thus potentially more logistically and financially feasible over the long-term than sipuleucel-T. [7]

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

demonstrated that the vaccine was able to generate a T-cell specific immune response and patients with the greatest magnitude of this not met its primary endpoint of overall survival in September 2017. Nonetheless, the combination of Prostvac and docetaxel remains response had superior outcomes. [10]. A phase III trial (NCT01322490) of Prostvac monotherapy, however, was reported to have scientifically rational and this trial will continue. Furthermore, at this point neither this trial nor the phase III trial have suggested a PROSTVAC has been investigated in 2 phase II trials in mCRPC, both of which administered the vaccine at monthly intervals until favor of PROSTVAC; the placebo was an empty poxviral vector containing no transgenes. As was seen in the sipuleucel-T studies, disease progression. An industry-sponsored, placebo-controlled, multicenter trial in 125 mCRPC patients randomized them 2:1 in patients receiving vaccine showed no change in TTP, yet had an overall survival benefit (25.1 months with PROSTVAC vs. 16.6 months with placebo; P = 0.0061). [6] (Figure 2) A second phase II study of PROSTVAC of 32 mCRPC patients at the NCI PROSTVAC is very well-tolerated, with common side effects of grade 1 injection-site reactions or flu-like symptoms. [9] safety concern for Prostvac.



Figure 1. Poxviral vaccine strategy. Modified poxvirus contains transgenes for the tumor-associated antigen PSA and 3 T-cell costimulatory molecules (TRICOM).

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC



Figure 2. PROSTVAC improved survival in mCRP patients in a randomized multi center phase II.

## 1.2.2 Rationale for Combining Vaccine with Docetaxel

docetaxel increased sensitivity to antigen-specific cytotoxic T cell killing and a broadening of the immune response resulting in the cancer cells. The resulting up-regulation of cell surface molecules like ICAM-1, MUC-1, and MHC class 1 molecules potentially enhancing immune recognition and immune mediated cell lysis by vaccine-activated immune cells. [11] Even non-lethal doses of vaccine. Docetaxel has been shown to induce immunogenic modulation resulting in changes in the surface antigen expression of There is important preclinical data that has been cultivated from studies in the LTIB supporting the combination of docetaxel and targeting of multiple antigens (antigen-cascade/spreading). [11, 12

#### Clinical Data

NCI clinical study. The phase II trial randomized 28 patients to docetaxel plus viral-vector based vaccine (vaccinia and fowlpox virus expressing PSA gene and the co-stimulatory gene B7.1) vs. vaccine alone. The combination was deemed safe; immune responses, as The clinical experience in prostate cancer utilizing the combination of chemotherapy and vaccines was previously investigated in an measured by antigen-specific-T cell activation against PSA antigen were equivalent in both arms suggesting that antigen specific Tcell activation at was unaffected by weekly docetaxel and the accompanying dexamethsone comedication. [9]

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

(TRICOM), similar to PROSTVAC. [13] This study randomized 48 patients to either docetaxel alone or docetaxel plus the PANVAC Additional data from a study involving breast cancer may have particular relevance in prostate cancer due to the use of docetaxel in vaccine. The final data suggested increased clinical benefit based on progression free survival (PFS) when vaccine was combined combination with PANVAC, a pox-viral vaccine, targeting MUC-1 and CEA and encoding three co-stimulatory molecules with docetaxel vs. docetaxel alone (PFS of 7.9 vs. 3.9 months, HR = 0.65, one-sided p=0.09).  $[\underline{14}]$  (Figure 3)



Figure 3. Comparison of progression-free survival (PFS). Medians: Docetaxel plus PANVAC vaccine 7.9 months versus docetaxel alone 3.9 months median PFS (p = 0.09, one-sided, meets predefined study statistical goal), HR = 0.65 (95% CI: 0.34 – 1.14). [14]

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

The combination of preclinical and clinical studies performed by our group here at the NCI provide a strong foundation for combining docetaxel and PROSTVAC in metastatic castration sensitive prostate cancer

# Initiating Therapies with Vaccines Earlier May Enhance Clinical Outcomes

cancer. (Tumor growth rates are based on tumor growth and regression kinetics and have been modeled using several relevant disease patients were on the therapy, but once the therapy became less effective or was discontinued, the growth rate reverted to pretreatment PROSTVAC, however, was not consistent with this previously demonstrated model. In this trial, no change in tumor growth rate was months. [10] However, unlike patients on chemotherapy, these patients' mortality could not be predicted by their post-treatment, offhave important implications. Using a mathematical equation to calculate tumor growth, survival can be predicted in several cancers cytoreductive therapies in other tumor types. Chemotherapy-based treatment temporarily altered or decreased the growth rate while rates and death was predictable based on the mathematical equation and off-study growth kinetics. [17] The vaccine trial involving study growth rates. Instead, these patients' survival times were more prolonged than would have been anticipated by their off-study patients with better vs. poor outcomes, suggesting that benefit from ensuing treatment does not account for this apparent disconnect including using disease-specific metrics, such as M-spike in multiple myeloma, tumor size in renal cell cancer and PSA in prostate Retrospective data from several studies suggests that therapeutic cancer vaccines may slow the growth rate of tumors and this can based on these growth rates. [17] When the 4 NCI trials that used cytotoxic were evaluated, the results were consistent with other growth rates. A separate analysis of this population indicated that subsequent therapies did not differentially improve survival for vaccine PROSTVAC, evaluated the impact of the various treatments on tumor growth rates and survival which can be calculated parameters. [15, 16] Using this equation, an analysis of 5 prostate cancer studies conducted at the NCI, including one using the seen while patients were on-study, consistent with that the trial had a median disease progression by conventional measures at between off-study growth rate and a far better survival time than would have been predicted using this model.

While this would be an unrealistic outcome with chemotherapy or hormonal therapy alone, given their transient clinical impact, it is One hypothesis regarding this outcome appears to be supported by data from other trials. Perhaps the tumor growth rate, which was plausible with immune therapies, which can initiate a persistent immune response that may evolve through antigen spreading well not significantly altered in the short term, was impacted in the time after treatment to such a degree that it improved survival. [18] beyond the treatment period. Other vaccine trials in prostate cancer have supported this hypothesis.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

These findings are consistent with the phenomenon of altered tumor growth kinetics following immune-based treatment, which affect trial of PROSTVAC in mCRPC all reported improved survival without changes in median disease progression frees survival. [6, 19] altering short-term disease progression, as evaluated by conventional measures such as PSA or RECIST-based imaging assessments. Indeed, multiple phase III trials of sipuleucel-T in mCRPC, a phase III trial of ipilimumab in metastatic melanoma, and the phase II In addition, larger clinical trials may support the hypothesis that some modern immune therapies alter tumor growth rate without long-term survival in the absence of any short-term decrease in tumor burden. If it is possible for therapeutic cancer vaccines to induce a dynamic and sustained immune response that indeed slows the growth rate of tumors, then it would appear rationale that initiating such an immune response earlier would have a greater impact than initiating that immune response later in the disease process.

This is one aspect of the new CHAARTED data that is so appealing. Six cycles of docetaxel with ADT improved survival by large impacting growth rate and having more impact on survival than has been seen in previous studies, where anticipated survival is magnitudes (greater than a year) over a 4-5 year timeline, providing the potential to enhance survival with immunotherapy by

## 1.2.4 Antigen Spreading/Antigen Cascade as an Endpoint

the immune response (i.e. more antigens being targeted) with improved clinical outcomes. [22-24] Based on these data, it is likely that response as they have the ability to be recognized by the immune system and will likely be present across multiple clonal populations cascade has been demonstrated in multiple studies and in multiple tumor types. Some studies have associated the greater breadth of Perhaps the greatest aspect of immunotherapy is its potential to induce an immune response that has the ability to evolve *in vivo*. [20] broader, adaptable, and personalized anti-tumor immune effect. As immunotherapies become more refined and immune monitoring When immune cells lyse cancer cells in the presence of an activated immune response, it is possible that additional antigens will be of cancer cells. It is then possible that when these secondary antigens are targeted and a subsequent population of cancer cells is initial immune target is not as important as the ability of initial immune response to lead to antigen cascade in vivo resulting in a taken up and processed by the immune system. These secondary antigen targets may be more relevant to the overall anti-tumor killed, additional antigens could be targeted in a similar manner.[21] This phenomenon known as antigen spreading or antigen

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

improves, it would seem that the breadth of immune response should be an important focus in the development of future immune strategies

treatment strategies have yet to be compared in prospective randomized trials and could inform future clinical trials with vaccines and It remains unclear whether vaccines combined with an immune stimulatory chemotherapy such as docetaxel enhances the immune associated immunosuppressive effects of the tumor have been diminished may also be a sound treatment strategy. [25] These two response more than sequential use. The use of vaccine after chemotherapy when the tumor has been cytoreduced and the volume other immunotherapies.

## 1.2.5 Evaluating Immune Response

markers of response, they have improved our knowledge of a vaccine-generated immune response and provided a better understanding of what factors are potentially important in mounting a sufficient anti-tumor immune response that could be associated with improved immunotherapy studies. A previous trial in mCRPC patients with PROSTVAC alone suggested that patients with greatest magnitude positioned and have the experience as the LTIB to conduct this rigorous immune testing from clinical samples of patients treated with clinical outcomes. These and other data have allowed us to optimize vaccines in subsequent clinical trials. Few groups are as well regulatory T-cell function were also associated with improved clinical outcomes. [26] While thethese findings are not surrogate of T-cell-specific response against PSA had favorable clinical outcomes. [10] That same trial also suggested that changes in Our group in the LTIB has previously evaluated immunologic parameters in clinical trials with PROSTVAC among several **PROSTVAC** 

### PSA-Specific Immune Responses

While many clinical trials have been done in biochemically recurrent prostate cancer, there is little reported on the impact of those therapies on the immunologic response that is near the depth and scope that is proposed in this trial. The proposed immunologic studies will be done on all patients by the Laboratory of Tumor Immunology and Biology at the NCI Clinical Center under the direction of Dr. Jeffrey Schlom

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

performed in biochemically recurrent prostate cancer patients. Advantages of this approach include the ability to assess both CD4 and Unlike previous studies involving PROSTVAC, which evaluated immune responses to a single 9 amino acid section of the 244 amino CD8 T cells, identification of multifunctional T cells (those producing  $\geq 2$  cytokines), and identification of T lymphocytes with lytic acid PSA protein, the immune analysis in this trial will evaluate overlapping 15 amino acid sequences of the entire PSA protein. PROSTVAC and a greater opportunity for clinical correlations. This type of analysis has not been previously prospectively (Figure 4). This more extensive analysis will provide a more thorough understanding of the immune response initiated by potential (CD107a expression). (Table 1).



Figure 4. Overlapping PSA Peptide Assessment. This innovative approach to evaluating for assessment of immune response to the entire PSA protein using overlapping 15 amin (Previous techniques have focused on assessing just one of these peptides.)




methods. (Responses are listed as absolute # of CD4 or CD8 T Lymphocytes Producing Cytokine or Positive for CD107a measured by CD107a expression. Had only one peptide been used to analyze this immune response it is likely that many Table 1. Preliminary Data from a Trial of PROSTVAC in mCRPC. This table shows how this multi peptide approach can be used in this proposal. In this previous (unpublished) trial, 2 cohorts of patients were evaluated using the proposed using multiple parameters (cytokine production signifying activation - IFN-y, IL-2 and TNF-a) and lytic potential as per 1x106 cells plated.) This readout shows the breadth of this analysis as both CD4 and CD8 tell cells are evaluated of these immune responders would not have been identified. (unpublished)

## Defining a Response and the Response Score

for CD4 or CD8 cells. For example, Patient #2 in Table 1 will be scored has having 5 responses (CD4: INFg, TNF and CD8: CD107a, A positive "response" will be defined as increased CD107a expression or increased intracellular cytokine production for given antigen INFg and TNF)

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

In order to give added weight to the spread antigens (MUC1 and Brachyury) they will be weighted 150% higher than PSA antigens. Thus the scoring will be as follows:

#### For PSA:

point each of the four CD4 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 4

1 point each of the four CD8 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 4

Total possible score for PSA response is 8

#### For MUC1:

1.5 points each of the four CD4 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 6

..5 points each of the four CD8 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 6

Total possible score for PSA response is 12.

#### For Brachyury:

1.5 points each of the four CD4 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 6

1.5 points each of the four CD8 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 6

Total possible score for PSA response is 12.

comparison will be made when combination therapy is complete in the docetaxel + PROSTVAC arm (19 weeks) and when sequential The primary comparison between the 2 arms will be at 19 weeks, with additional comparisons at 39 weeks and 1 year. In addition, a therapy is stopped in the docetaxel followed by PROSTVAC arm (39 weeks).

# 1.2.6 Flow Cytometry Analysis of Immune subsets (Biomarker Development)

prior to therapy. The score is calculated from the changes in frequency of certain immune cell subsets after vaccine treatment. The develop a Peripheral Immunoscore based on the frequency of specific pre-determined immune cell subsets in the blood of patients subsets. (Table 2). This methodology has been previously described (13). This added analysis will provide preliminary data to As part of the extensive immune interrogation, peripheral immune cells will be evaluated by 30 markers to assess 127 immune resultant panel of markers would reflect immune response to the vaccine.

## Table 2. Analysis of Peripheral Immune Cells

- 1. **CD4**: Helper T lymphocytes (32 subsets)
- 2. **CD8**: Cytotoxic T lymphocytes (29 subsets)

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- Markers of PD-1 pathway and T cell activation (in CD4 and CD8):
  - **EOMES:** activation
- TCR-αβ: activation
- Tbet: activation
- **BATF:** activation/exhaustion
- Maturation status of T lymphocytes (in CD4 and CD8):
  - Naïve: CD45RA<sup>+</sup> CCR7<sup>+</sup>
- Effector Memory: CD45RA- CCR7-
- Ferminal (EMRA): CD45RA+ CCR7-
- Tlymphocyte markers (in CD4 and CD8):
- CTLA-4: inhibition
- PD-1: activation/inhibition
- PD-L1: activation/cross-inhibition
- TIM-3: inhibition
- ICOS: activation (only on CD4)
- **Tregs**: Regulatory T lymphocytes (CD4<sup>+</sup> CD25<sup>+</sup> FoxP3<sup>+</sup> CD127<sup>-</sup>) (7 subsets)
- CD45RA: Tregs highly expandable in vitro
- CTLA-4: Treg suppression
- CD49d: "contaminating" effector lymphocytes (non-Tregs)
- ICOS: Treg suppression
- PD-1: activation/inhibition PD-L1: cross-inhibition
- **B lymphocytes**: CD19<sup>+</sup> (5 subsets)
  - CTLA-4: inhibition

  - TIM-3: inhibition
- PD-1: activation/inhibition
- PD-L1: cross-inhibition
- NK: Natural killer cells (CD56<sup>+</sup> CD3<sup>-</sup>) (20 subsets) 5.
- CD16+ CD56br: Functional intermediate, lytic and cytokine production
  - CD16+ CD56dim: Mature NK, cytokine production
- CD16- CD56br: Immature, abundant in human placenta
  - CD16 CD56dim: non-lytic, non-cytokine production
- PD-1: activation/inhibition

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- **PD-L1:** cross-inhibition
- 6. **NK-T**: CD56<sup>+</sup> CD3<sup>+</sup> (4 subsets)
- TIM-3: activation
- **PD-1:** activation/inhibition
- **PD-L1:** cross-inhibition
- cDCs (Conventional DCs): CD3-CD56-CD1c+CD303- (5 subsets)
- pDCs (plasmacytoid DCs): CD3-CD56-CD1c-CD303+ (5 subsets)
- Markers of DC activation
- CD83: activation
- TIM-3: inhibition
- **PD-1:** activation/inhibition
- **PD-L1:** cross-inhibition
- 9. **MDSCs**: Myeloid-derived suppressor cells (CD11b<sup>+</sup> HLA-DR<sup>low/-</sup>CD33<sup>+</sup>) (20 subsets)
- CD14: Common Myeloid Marker (high in monocytes, dim in granulocytes)
- CD15: Granulocyte marker
- CD16: most immature monocytic MDSCs
- **PD-1:** activation/inhibition
- **PD-L1:** cross-inhibition

### 1.2.7 Pharmacogenomic Studies

genes involved in facilitation of drug transporters, 9 genes involved in global regulation of drug metabolizing/transporting proteins, 4 assess genotype of the most relevant drug metabolizing enzymes and transporters (DMET). DNA will be analyzed on a DMET Plus metabolism) genes, 13 non-CYP (phase I metabolism) genes, 78 phase II metabolizing genes (including UGTs), 63 transporters, 4 One blood sample per patient will be collected in a purple top tube for pharmacogenetic studies to analyze the genomic DNA and (Affymatrix) genotyping platform that tests for 1,936 genetic variations in 225 drug disposition genes, including 47 CYP (phase I drug binding proteins, and 4 drug targets.

which are included in the DMET analysis. OATP1B3 genotype is particularly interesting based on a previous study that demonstrated a polymorphism that is predictive of response to ADT therapy failure. [27] Men with at least one copy of the wild-type allele (T) at Of specific interest to DTX are polymorphisms in CYP3A4/5 (metabolism), ABCB1 (transport), and OATP1B3 (transport), all of

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

position 334 have a shorter time (p=0.048) from ADT to AI (1.2 yrs) versus men with two copies of the mutant (G) allele (1.57 yrs), consistent with in vitro data that the wild-type SLCO1B3 is more functional at importing testosterone vs the mutant (G-allele) [28]. Experimental Imaging May Help improve our understanding of castration sensitive disease progressing to castration resistant 1.2.8

rapidly advancing the field of radiology. In collaboration with the NCI's Molecular Imaging Program under the direction of Dr. Peter which have been used to evaluate prostate cancer for nearly 3 decades, but the field has not benefited from newer technology that is Choyke, several experimental and emerging imaging platforms will be evaluated with the ultimate goal of prospectively evaluating Conventional imaging in prostate cancer primarily consists of computed tomography (CT) scans and technetium-99m bone scans, these tools both individually and in combination as a means to assess castration sensitive disease and its ultimate progression to castration resistant disease. Each platform has a sound rationale for its use in this population and are detailed below.

radiation therapy) or in the prostate bed (in the case of radical prostatectomy). Typically, the latter are found around the urethra, often **Endorectal MRI:** For local recurrence or locally untreated prostate cancer, the preferred method is multiparametric MRI typically enhanced (DCE) MRI. Recurrences typically enhance early and more profoundly than surrounding tissue. Because MRI does not near the anastomosis. These are detected with high resolution MRI particularly employing T2 weighted and dynamic contrast with an endorectal coil at 3T. MRI has the ability to localize small deposits of disease within the prostate (in the case of prior involve radiation it is highly amenable to repeated scanning for therapeutic monitoring.

limitation of its use in monitoring bone metastases is that there can be a "lagging indicator" of response. Despite response to therapy, substantially faster than conventional bone scan (can be performed within 1 hour of injection) sodium fluoride PET/CT has the added degenerative changes on CT, eliminating them further consideration. Software is now available to automatically detect true positive Sodium Fluoride (NaF) PET: For advanced disease, sodium fluoride PET is the most sensitive method of detecting prostate cancer osteoblastic bone metastases. [29, 30] (Figure 5) Sodium fluoride is incorporated into the bone matrix. Thus during osteoblastic bone sodium fluoride images, which can then be monitored over time. Increases in standardized uptake value (SUV) are associated with Sodium fluoride PET/CT has proven to be substantially more sensitive than conventional Tc-99m bone scans. In addition to being formation, there is avid uptake of the radiolabeled agent. Very small doses (3mCi) of activity are needed for satisfactory imaging. progressive disease. Thus, sodium fluoride PET/CT is the most sensitive method to detect prostate cancer bone metastases. One virtue of providing a registered CT scan to the PET image. Many lesions identified on the PET scan can be correlated with

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

some bone metastases continue to show activity on sodium fluoride PET/CT due to the ongoing osteoblastic remodeling. For this reason, substantial changes in SUV are required before one can conclude that disease is progressing or regressing on NaF scans.

#### 1.2.9 Rationale for Arm C

chemotherapy and determine if that would be an optimal sequence. Certainly an activated immune response prior to cytotoxic therapy second). This was largely due to the fact that we did not anticipate having patients contact us who recently started ADT. In fact, the majority of patients enrolled on this study started ADT under our care or direction. Thus, since the standard therapy for this regimen is to initiate ADT and then subsequently start chemotherapy within 4 months, it provided an opportunity to initiate vaccine prior to unknown in medical oncology. The trial was originally designed to answer the question of concurrent vs. sequential (with vaccine The primary goal of this clinical trial is to evaluate the optimal timing of immunotherapy with chemotherapy as this is largely could synergize with the chemotherapy as supported by preclinical data above (section 1.2.2), but we do not have clinical/immunologic data on this from human studies. This study can provide to address this scientific question,

primary endpoints are immunologic and will be assessed at the end of the study, they cannot be influenced by provider knowledge of a Given that Arm A and B have nearly completed accrual, we are unable to randomize patients among all 3 Arms. Thus Arm C will be assignment as much as possible and that is why more patients are required (26 vs. 17). Regardless, this comparison would Arm C to need to be taken into account with any analysis done. Regardless, the nature of this study would require a future confirmatory study. Arm A and B will provide valuable insight into optimal sequencing of immunotherapy with chemotherapy. Furthermore, since the non-randomized arm. It is possible that patient variations may exist between Arm A or B vs. Arm C, but that is something that will for patients who have started ADT within 1 month of enrollment. The statistical design compensates for the lack of random




in a patient whose bone scan was negative will allow for a composite assessment that findings. This proposal will prospectively remains undefined. Patients evaluated as Figure 5. Increase Sensitivity of <sup>18</sup>F-NaF increased sensitivity of <sup>18</sup>F-NaF PET/CT biochemically recurrent prostate cancer imaging confirms findings such as these after longer follow-up. In addition, the use of multiple radiographic platforms part of this proposal will be followed prospective value of such findings in could improve the specificity of such prospectively to see if conventional PET/CT. This case illustrates the but PET/CT was positive. The

## ELIGIBILITY ASSESSMENT AND ENROLLMENT

### 2.1 ELIGIBILITY CRITERIA

- 2.1.1 Inclusion Criteria
- 2.1.1.1 Documented histopathological confirmation of prostate cancer from a CLIA-certified laboratory.
- Patients must have metastatic disease, defined as at least one lesion on bone scan or at least one lesion that are measurable per RECIST 1.1 (see section 6.3.2). (Patients who have metastatic disease by these criteria prior to ADT, but then have changes after ADT that diminish the size of these lesions or changes on bone scan are still eligible.)
- Patients must have a performance status of 0 to 2 according to the ECOG criteria (see Appendix B)
- 2.1.1.4 Patients must have adequate bone marrow, hepatic, and renal function with:
- ANC  $\geq 1500/\mu$ L, without CSF support
- Platelets  $\geq 100,000/\mu L$

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- AST(SGOT)  $\leq$  2.5 x upper limit of normal (ULN);
- ALT(SGPT)  $\leq$  2.5 x upper limit of normal (ULN);
- Total serum bilirubin  $\leq 1.5$  x upper limit of normal (ULN), OR in patients with Gilbert's syndrome, a total bilirubin  $\leq 3.0$ )
- Serum albumin  $\geq 2.8 \text{ g/dL}$
- Lipase < 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis
- Creatinine  $\leq 1.5 \text{ X}$  institutional upper limits of normal

OR

 $\geq$  50 ml/min/1.73 m2 for patients with creatinine levels above institutional normal by 24-hour Creatinine clearance of urine.

- 1.1.5 Willing to travel to the NIH for follow-up visits
- 2.1.1.6 18 years of age or older.
- .1.1.7 Able to understand and sign informed consent.
- May have had up to 24 months of ADT (testosterone suppression therapy) in the nonmetastatic setting and are at least 12 nonths removed from treatment. 2.1.1.8
- Men treated or enrolled on this protocol must also agree to use adequate contraception, prior to the study, for the duration of months after the last dose of study drug(s). Should a woman become pregnant or suspect she is pregnant while her partner is medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 must also agree to use both a barrier method and a second method of birth control during the course on the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential study participation, and 4 months after completion. Sexually active subjects and their female partners must agree to use participating in this study, she should inform her treating physician immediately. 2.1.1.9
- 2.1.1.10 Must have started ADT for metastatic disease within 134 days (for Arm A and B) or within 30 days (for Arm C).

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- 2.1.2 Exclusion Criteria
- 2.1.2.1 Immunocompromised status due to:
- Human immunodeficiency virus (HIV) positivity.
- Active autoimmune diseases such as Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjögren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome or active Grave's disease. Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including CNS, heart, lungs, kidneys, skin, and GI tract will be allowed.
- Other immunodeficiency diseases
- by investigator within 28 days before the first planned dose of PROSTVAC. Use of inhaled steroids, nasal sprays, and topical Chronic administration (defined as daily or every other day for continued use > 14 days) of corticosteroids deemed systemic creams for small body areas is allowed.
- 1.2.3 Evidence of rising PSA on ADT
- Serious intercurrent medical illness that, in the judgment of the investigator, would interfere with patient's ability to carry out he treatment program.
- Other medications used for urinary symptoms including 5-alpha reductase inhibitors (finasteride and dutasteride) and alternative medications known to alter PSA (e.g. phytoestrogens and saw palmetto) 2.1.2.5
- History of allergic reactions attributed to compounds of similar chemical or biologic composition to poxviral vaccines (e.g., /accinia vaccine) 2.1.2.6
- Known allergy to eggs, egg products, aminoglycoside antibiotics (for example, gentamicin or tobramycin).
- History of atopic dermatitis or active skin condition (acute, chronic, exfoliative) that disrupts the epidermis
- 2.1.2.9 Previous serious adverse reactions to smallpox vaccination
- vaccination: (a) children  $\leq 3$  years of age, (b) pregnant or nursing women, (c) individuals with prior or concurrent extensive 2.1.2.10 Unable to avoid close contact or household contact with the following high-risk individuals for three weeks after the Day 1 eczema or other eczemoid skin disorders, or (d) immunocompromised individuals, such as those with HIV.
- 2.1.2.11 Receipt of an investigational agent within 28 days (or 60 days for an antibody-based therapy) before the first planned dose of

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- 2.1.2.12 Patients who test positive for HBV or HCV
- 2.1.2.13 Uncontrolled hypertension (SBP>170/ DBP>105)
- 2.1.2.14 Patients who have had prior chemotherapy for prostate cancer.
- 2.1.2.15 The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic reatment (with the exception of nonmelanoma skin cancers or carcinoma in situ of the bladder).
- 2.1.2.16 The subject has active brain metastases or epidural disease.
- 2.1.2.17 Patients with greater than or equal to grade 2 peripheral neuropathy at baseline.
- 2.1.2.18 Patients with history of splenectomy.

### 2.1.3 Recruitment Strategies

This study will be listed on available websites (www.clinicaltrials.gov, https://ccr.cancer.gov/clinical-trials-search-start) and participants will be recruited from the current patient population at NIH.

### 2.2 SCREENING EVALUATION

- A. Pathological confirmation of diagnosis by a CLIA certified laboratory may be obtained any time prior to enrollment.
- B. The following parameters will be obtained within 8 weeks prior to start of treatment:
- HIV test
- Hepatitis B and C
- Tc-99 whole-body scintigraphy
- CT (or MRI may be substituted at investigator's discretion) of chest, abdomen and pelvis
- History and physical examination including vital signs
- ECOG performance status
- Complete blood count plus differential and platelet count
- Hepatic (alkaline phosphatase, AST, ALT, total bilirubin, direct bilirubin), Mineral (albumin, calcium, magnesium, phosphorus) and Acute Care (sodium, potassium, chloride, bicarbonate, creatinine, glucose, BUN, eGFR) Panels
- Serum lipas

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- Serum PSA
- Testosterone level

### .3 BASELINE EVALUATION

To be performed within 16 days prior start of treatment (these tests will not need to be repeated if they were done at screening within the appropriate timeframe):

- History and physical exam including weight and vital signs
- ECOG performance status
- CBC with differential and platelet count, prothrombin time/INR, activated partial thromboplastin time
- Urinalysis (may be omitted in patients with incontinence who cannot produce a clean sample)
- Serum chemistries (Na+, K+, Cl-, CO2, BUN, creatinine, glucose, AST/ALT, bilirubin, calcium, phosphorous, albumin, magnesium, alkaline phosphatase, LDH, ionized calcium, amylase, lipase, total protein, GGT, uric acid)
- Serum Testosterone level
- Serum PSA
- Lymphocyte phenotyping CD3/CD4/CD8
- Baseline electrocardiogram 12 lead ECG (EKG) on all patients, and appropriate cardiologic evaluation, as clinically indicated, to provide baseline function and identify any patients who should be monitored closely for cardiac risks associated with vaccinia vaccination
- HLA-A, B, C and HLA-A\*02 and A\*03 subtype may be collected at any time during the study if not previously collected. This test does not need to be repeated prior to enrollment if previously collected at NIH.
- Biopsy (optional)
- Endorectal MRI (optional)

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## ..4 REGISTRATION PROCEDURES

ncicentralregistration-l@mail.nih.gov. After confirmation of eligibility at Central Registration Office, CRO staff will call pharmacy to with NCI Central Registration Office (CRO) within 24 hours of signing consent. To initially register a subject after the participant has Registration will be a two-part process as patients are screened on this protocol. Authorized staff must register an eligible candidate (http://home.ccr.cancer.gov/intra/eligibility/welcome.htm) indicating that the patient is being registered for screening and send via completion of screening studies, complete the remainder of the form which is the eligibility checklist, indicating that the patient is Registration will be forwarded electronically via e-mail to the research team. A recorder is available during non-working hours. encrypted email to: NCI Central Registration Office ncicentralregistration-l@mail.nih.gov. Once eligibility is confirmed after advise them of the acceptance of the patient on the protocol prior to the release of any investigational agents. Verification of being registered for treatment and fax the completed registration checklist to the CRO at NCI Central Registration Office signed the consent, complete the top portion the registration Eligibility Checklist from the website

Subjects that do not meet screening criteria should be removed from the study following the procedure in section 3.3.3.

# 2.4.1 Treatment Assignment and Randomization/StratificationProcedures

#### Cohorts

| Number Name | Name | Description |
|---|---|---|
| 1 | ADT established | Patients who have started ADT for metastatic prostate cancer no more than 134 days prior and no fewer than 29 days prior to enrollment |
| 2 | ADT not yet established | ADT not yet established Patients who have not started ADT or who have been on ADT for 28 days or fewer |

#### Arms

| Letter | Name | Description |
|---|---|---|
| A | Sequential docetaxel followed by | 6 cycles of docetaxel followed by PROSTVAC |

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

| | <u>PROSTVAC</u> | |
|---|---|---|
| В | Combined docetaxel with PROSTVAC | 6 cycles of docetaxel concurrently administered with PROSTVAC |
| C | PROSTVAC prior to docetaxel | 4-6 injections of PROSTVAC followed by 6 cycles docetaxel |

#### Stratifications

| Name | Distinct Options | Notes |
|---|---|---|
| Disease Volume | High<br>Low | Done at time of randomization to minimize differences n disease volumes between arms |

## Randomization and Arm Assignment

Subjects in Cohort 1 will be stratified and randomized on a 1:1 basis between Arm A and Arm B. The computerized randomization will be performed by the Central Registration Office.

Subjects in cohort 2 will be directly assigned to Arm C.

CRO staff will send a secured e-mail to Principal Investigator and research nurse with the Verification of Registration of the patient and treatment arm patient is randomized. This process will be completed within 15-30 minutes of faxing the eligibility checklist. CRO will keep track of all randomization data in Clinical Data Registry (CDR) of CRO.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## STUDY IMPLEMENTATION

#### 3.1 STUDY DESIGN

cycles (Arm B) versus ADT followed by sequential docetaxel 75 mg/m2 q3 weeks x 6 cycles followed by PROSTVAC q3 weeks x 6 This is a randomized trial of ADT followed by simultaneous docetaxel 75 mg/m2 q3 weeks x 6 cycles + PROSTVAC q3 weeks x 6 cycles (Arm A) in men with newly diagnosed mCSPC.

after week 9 or with confirmed rise in PSA based on investigator discretion. After vaccine discontinuation, docetaxel will be initiated vaccinia-PROSTVAC 2x10<sup>8</sup> infectious units subcutaneously will be initiated within 28 days of starting ADT. This will be followed within 28 days of last vaccine but not beyond 134 days of initiating ADT. Docetaxel will be given alone at 75 mg/m<sup>2</sup> intravenously by fowlpox-PROSTVAC booster 1x10<sup>9</sup> infectious units subcutaneously on weeks 3, 6, 9, 12 and 15. Vaccine may be discontinued Arm C will evaluate patients who have not started ADT or who have been on ADT for no more than 28 days. For these patients, every three weeks for a total of 6 doses.

### 3.1.1 Protocol Stopping Rules

- This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for grading systemic
- One occurrence of grade 5 toxicity by the NCI-CTCAE version 4.0 attributable to the treatment regimen.
- Two occurrences of grade 4 toxicity by the NCI-CTCAE version 4.0 attributable to the treatment regimen

### .2 DRUG ADMINISTRATION

#### 2.1 AD7

Standard ADT will be used based on standard dosing scheduling. GnRH agonists and GnRH antagonist are acceptable as long as patients maintain castrate levels of testosterone. Orchiectomy would also be an option if that is desired by the patient.

### 3.2.2 PROSTVAC Vaccine

All vaccines in this trial should be handled according to the guidelines outlined by each department. Study staff administering the department or unit. Patients receiving PROSTVAC-V should be isolated just prior to the administration of vaccine and can be vaccine or assessing the vaccine site should wear personal protection consistent with the standard of practice outlined by each

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

removed from isolation after the vaccine is administered and bandage is secured over the injection site. Appendix C defines individuals at risk for vaccinia exposure.

## 3.2.2.1 Arm A – sequential docetaxel + PROSTVAC

PROSTVAC-V (vaccinia) will be administered subcutaneously in week 19 at a dose of 2x10<sup>8</sup> infectious units.

PROSTVAC-F (fowlpox) will be administered subcutaneously at a dose of 1x10<sup>9</sup> infectious units starting in week 21. Administration on day 1 of each cycle will continue for 6 cycles. (Weeks 21, 24, 27, 30, 33 and 36)

## 3.2.2.2 Arm B – concurrent docetaxel + PROSTVAC

PROSTVAC-V (vaccinia) will be administered subcutaneously in week -2 at a dose of 2x10<sup>8</sup> infectious units.

PROSTVAC-F (fowlpox) will be administered subcutaneously at a dose of 1x109 infectious units starting on day 1, week 1. Administration on day 1 of each cycle will continue for 6 cycles. (Weeks 1, 4, 7, 10, 13 and 16)

## 3.2.2.3 Arm C - PROSTVAC prior to Docetaxel

PROSTVAC-V (vaccinia) will be administered subcutaneously in week 1 at a dose of 2x108 infectious units.

PROSTVAC-F (fowlpox) will be administered subcutaneously at a dose of 1x109 infectious units starting on week 3. Administration on day 1 of each cycle will continue for 5 total cycles. (including Weeks 6, 9, 12, 15). Vaccine may be discontinued after week 9 or with confirmed rise in PSA based on investigator discretion at which time docetaxel could begin within 28 days. One dose of vaccinia-PROSTVAC and 3 doses of fowlpox-PROSTVAC may be adequate to generate an immune response based on previous studies. The investigator may use clinical discretion to forgo dose 4 and 5 of fowlpox-PROSTVAC and initiate chemotherapy.[10] In addition, for patients who may have a rise in PSA while on vaccine alone, vaccine can be discontinued early at the discretion of the investigator and docetaxel can be initiated with confirmed rise in PSA.

#### 3.2.2.4 Dosing Delay

Patients must have recovered to ≤ grade 1 toxicity related to vaccine for the parameters used to assess levels of organ function required for eligibility (see Section 2.1) after each vaccination in order to receive a subsequent vaccination.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- If  $\geq$  grade 3 nonautoimmune toxicity attributable to the vaccine persists for > 42 days, the patient will not receive further vaccine inoculations and will be removed from the protocol treatment and followed for resolution of toxicity and immune/survival endpoints.
- Patients who develop grade 3 injection site reactions will have their vaccine held until injection site reaction resolves to grade 2 or less.
- Patients who develop  $\geq$  a grade 2 allergic or autoimmune disease that threatens vital organ function or any  $\geq$  grade autoimmunity, not related to a therapeutic response, will be removed from the protocol treatment and followed for resolution of toxicity and immune/survival endpoints.
- Patients who develop any grade 4 toxicity attributable to vaccine will be removed from the protocol treatment and followed for resolution of toxicity and immune/survival endpoints.
- If a scheduled vaccine or docetaxel dose is missed due to scheduling or logistical issues, the vaccine or docetaxel may be given within 7 days of the appointed time.

### 3.2.2.5 Dose modifications

No dose modifications are allowed with this vaccine.

#### 3.2.3 Docetaxel

Appropriate dose modifications are described. No investigational or commercial agents or therapies other than those described may be Treatment will be administered primarily on an outpatient basis. Reported adverse events and potential risks are described. administered with the intent to treat the patient's malignancy.

| Agent | Premedications Dose | | Route | Route Schedule Cycle | Cycle |
|---|---|---|---|---|---|
| | | | | | length |
| Docetaxel | 8 mg of oral | <i>SL</i> | IV over 1 | IV over 1 Day 1 for 21 days | 21 days |
| | dexamethasone | mg/m2 | hour | Arm A | (3 weeks) |
| | 12 hours, 3 | | | | |
| | hours, and 1 | | | Day 2 or | |
| | hour before | | | Day 3 for | |
| | infusion <b>OR</b> | | | Arm B | |
| | 12 mg IV 15- | | | | |

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

| 30 minutes |
|---------------------------------------|
| prior to |
| · |
| infusion |

Docetaxel 75mg/m² will be administered intravenously as described in Appendix D every 21 days (i.e., a 3-week cycle) for up to 6 cycles. All patients will receive 8 mg of dexamethasone orally 12 hours, 3 hours and 1 hour prior to docetaxel infusion OR may receive dexamethasone 12 mg intravenously prior to docetaxel.

In the event of a hypersensitivity reaction, infusion times may be longer. Hypersensitivity reactions may be managed clinically according to PI discretion. Please see Appendix D for suggested management guidelines (optional). To minimize patient exposure to phthalate plasticizers (e.g., DEHP), which may be leached from PVC containers and administration sets, administer docetaxel only through polyethylene-lined administration sets.

#### 3.2.3.1 Dose Reduction

| Dose Level | Docetaxel (mg/m <sup>2</sup> ) |
|------------|--------------------------------|
| Level 0 | 75 mg/m <sup>2</sup> |
| Level - 1 | 65 mg/m <sup>2</sup> |
| Level - 2 | 55 mg/m <sup>2</sup> |

## 3.2.3.2 Docetaxel Dose Modifications

Patients should have an ANC  $\geq$ 1500 cells/mm<sup>3</sup>, a platelet count  $\geq$  75,000 cells/mm<sup>3</sup> (grade 1 hematologic toxicity) and resolution of any grade 3 or higher non-hematologic toxicity to < grade 1 or baseline in order to initiate another treatment cycle of docetaxel For febrile neutropenia developed within a prior cycle, docetaxel can be continued during future cycles at a dose reduction d and if patients will be treated with filgrastim support. Docetaxel will be resumed at the same dose once neutropenia has resolved to  $\leq$  grade indicated, with the addition of filgrastim support. For grade 4 neutropenia lasting greater than 5 days docetaxel will be held and

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## Docetaxel Dose Modifications for Neutropenia without Fever:

| When Neutrophils fall to | for a Duration<br>of | for a Duration Recommended Course of |
|---|---|---|
| <1000 but \ge 500/mcL (Grade 3) | Any length of time | $<1000$ but $\geq 500$ /mcL (Grade Any length of No dose reduction for future cycles. 3) |
| <500/mcL (Grade 4) | <pre>&lt; 5days</pre> | No dose reduction for future cycles. |
| <500/mcL (Grade 4) | > 5 days | No dose reduction. DOCETAXEL will be held and patients will be treated with filgrastim support. DOCETAXEL will be resumed at the same dose once neutropenia has resolved to ≤ grade 1 or baseline. |

For grade 3 constipation or grade 3 fatigue, treatment can resume with a dose reduction after resolution of toxicity to  $\leq$  grade 1 or baseline. Study Calendar

See Appendix A.

# 3.3 CRITERIA FOR REMOVAL FROM PROTOCOL THERAPY AND OFF STUDY CRITERIA

Prior to documenting removal from study, effort must be made to have all subjects complete a safety visit within 30 days following the last dose of study therapy (see section 3.4).

## 3.3.1 Criteria for removal from protocol therapy

Patients will be removed from treatment for the following:

- Clinical or radiographic progression of disease.
- Serological progression, as defined in protocol section 6.3.6, may remain on treatment at the discretion of the PI.
- Grade 2 or greater autoimmune disease that threatens vital organs (Patients may be given the option to continue the study with standard of care docetaxel as clinically indicated with no further vaccine),
  - Grade 3 or greater autoimmune response that is not related to a therapeutic response (Patients may be given the option to continue the study with standard of care docetaxel as clinically indicated with no further vaccine).

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- Any Grade 4 non-heme toxicity that is possibly, probably or definitely related to the protocol treatment will require a patient to be off-treatment.
- Intercurrent illness or medical circumstances. If at any time the constraints of this protocol are detrimental to the patient's health, the patient may be removed from protocol therapy and reasons for withdrawal will be documented.
- Any grade of seizure will require a patient to be off-treatment.
- Completion of protocol therapy.

#### 3.3.2 Off-Study Criteria

- Patient is off-treatment and/or has agreed to be followed on a long term therapy protocol as outlined in section 3.5.
- Patient requests to be taken off study. Reasons for withdrawal will be documented
- Noncompliance with protocol guidelines (patient removed at discretion of Principal Investigator).
- Death
- Screen failure

## 3.3.3 Off Protocol Therapy and Off-Study Procedure

taken off-study. A Participant Status Updates Form from the web site (http://home.ccr.cancer.gov/intra/eligibility/welcome.htm) main Authorized staff must notify Central Registration Office (CRO) when a subject is taken off protocol therapy and when a subject is page must be completed and sent via encrypted email to: NCI Central Registration Office ncicentralregistration-l@mail.nih.gov

### 3.4 FOLLOW-UP EVALUATIONS

safety visit within 30 days of drug discontinuation. The safety assessments may be performed by a local physician and laboratory if patients are unable to return to the NIH Clinical Center at this time. The investigator will contact the local physician to discuss the After subjects have stopped taking the study medication for any of the reasons listed in Section 3.3, they will be seen at NIH for a safety assessments outlined below and request that medical records be sent to the NIH. Patients who completed protocol therapy including the safety visit without disease progression will be followed every 12 weeks +/- 6 weeks until disease progression. Disease progression is defined in Section 6.3.

The following assessments will be performed during the follow up and safety visit:

- History and Physical Examination
- CBC with differential and platelet count, prothrombin time/INR, activated partial thromboplastin time

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- Serum chemistries (Na+, K+, Cl-, CO2, BUN, creatinine, glucose, AST/ALT, bilirubin, calcium, phosphorous, albumin, magnesium, alkaline phosphatase, LDH, ionized calcium, amylase, lipase, total protein, GGT, uric acid)
- Serum PSA level
- Adverse event reporting as needed as defined in section 7.

term therapy protocol as outlined in section 3.5 to find out how they are doing and to determine survival status. If there are unresolved During the safety visit, if there are no unresolved grade 3 or higher AEs, we may, when feasible ask the patient to enroll on the long grade 3 – 4 AEs, patients will be followed either at the NIH Clinical Center or by their local physician. In the latter case, we will obtain the physician's record of AEs.

Any scans performed outside of the NIH will also be obtained when possible.

### 3.5 POST-STUDY EVALUATION

Information regarding the findings will be reported to the FDA. Patients assigned to receive PROSTVAC will be offered enrollment in The Biologic Response Modifiers Advisory Committee has recommended that long-term follow-up extend over a period of 15 years. the 04-C-0274 "Follow-Up Study of Subjects Previously Enrolled in Immunotherapy Studies Utilizing Gene Transfer or other immunotherapeutic agents" once off study.

## CONCOMITANT MEDICATIONS/MEASURES

Subjects must inform the investigators of the current or planned use or all other medications during the study (including prescription medications, vitamins, herbal and nutritional supplements, and over-the-counter medications). For the administration of PROSTVAC, antiemetics, stool softeners and antidiarrheal agents may be administered as required, but are not anticipated to be needed and should not be used prophylactically on the first cycle. The selection of the specific antiemetic regimen is at the discretion of the treating physician. Antiemetic regimens will not include steroids. Other supportive care with blood components, antibiotics, analgesics, general medical therapy, etc., will be delivered as required. Any patients taking antibiotics for any reason must complete that course of therapy and be free of evidence of further infection before receiving any dose of vaccine. Concurrent systemic corticosteroid use (daily or every other day for continued use > 14 days) should be avoided within 28 days before the first planned dose of PROSTVAC. Use of inhaled steroids, nasal sprays, and topical creams for small body areas is allowed.

Symptomatic anemia should be treated with appropriate red blood cell or erythropoietin support.
Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Thrombocytopenia should be treated conservatively. In the absence of bleeding or a planned invasive procedure, platelet transfusions should be given for a platelet count below 10,000/mm3. If invasive procedures are planned or the patient develops bleeding, platelet transfusions should be administered in accordance with the standard of practice, usually maintaining a platelet count of > 50,000/mm3.

Any evidence of disseminated intravascular coagulation (DIC), hemolytic uremic syndrome (HUS), or thrombotic thrombocytopenic purpura (TTP) including thrombocytopenia, hemolytic anemia, renal failure, fever or neurologic changes should be thoroughly evaluated and closely monitored and supported as clinically indicated.

# 4.1 CONCURRENT MEDICATIONS/INTERVENTIONS

### 4.1.1 Anticancer Therapy

If a subject requires additional systemic anticancer treatment, study treatment must be discontinued. Local intervention is discouraged unless medically unavoidable. Subjects receiving local intervention (e.g., palliative radiation) are allowed to continue to receive study treatment at the investigator's discretion.

### 1.1.2 Other Medications

(including prescription medications, over-the-counter medications, vitamins and herbal and nutritional supplements). It is the Subjects must be instructed to inform the investigators of the current or planned use or all other medications during the study responsibility of the investigator to ensure that details regarding all medications are documented. Bisphosphonates started prior to screening activities or initiated during the course of the study to control bone pain may be used with caution. Colony stimulating factors (e.g., erythropoietin and granulocyte colony-stimulating factors) administered as dictated by safety purposes are acceptable while the subject is enrolled on study. Pain medications administered as dictated by standard practice are acceptable while the patient is enrolled on the study.

No concurrent investigational agents are permitted

#### 4.1.3 Neutropenia

Growth factors may be used as medically indicated if patient develops fever and neutropenia. Dose reduction or interruption of docetaxel is also recommended as described.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 4.2 TREATMENT OF VACCINIA VACCINATION COMPLICATIONS

## 4.2.1 Vaccinia Immune Globulin (VIG)

and progressive vaccinia) is with VIG. VIG is contraindicated, however, for the treatment of isolated vaccinial keratitis. VIG is a inoculation involving extensive lesions or if comorbid conditions exist, severe cases of generalized vaccinia in patients that are sterile solution of the immunoglobulin fraction of pooled plasma from individuals inoculated with vaccinia vaccine. VIG is only available through the CDC's Strategic National Pharmaceutical Stockpile by contacting the CDC's Clinician Information Line at 1-877-554-4625 or the Director's Emergency Operations Center (DEOC) at 770-488-7100. Upon receipt of a call from a patient or upon direct observation of a patient, or contact, who manifests signs and symptoms of any of the above conditions, the investigator should First-line treatment of some of the complications of vaccinia caused by dissemination of vaccinia virus (severe cases of inadvertent systemically ill and whose condition might be toxic or who have serious underlying immunosuppressive illnesses, eczema vaccinatum, place a call to the CDC as soon as possible:

- 1) to initiate review of the clinical case,
- 2) to seek consultation on the appropriateness of VIG therapy,
- 3) to determine the appropriate VIG dose and dosing method for administration, if VIG therapy is required, and
- 4) to determine how to access and have the appropriate doses of VIG delivered.

is contraindicated for treatment of isolated vaccinial keratitis due to the increased risk of corneal scarring. A new IV formulation of Early institution of VIG therapy is advised following recognition of clinical symptoms compatible with some vaccinia complications (eczema vaccinatum, severe generalized vaccinia, progressive vaccinia, and some cases of inadvertent inoculation). The effectiveness VIG that has a lower level of aggregated protein allowing it to be used by either the IM or IV route is available through the CDC. This formulation will most likely be preferred for administration and the CDC will instruct investigators regarding appropriate dosing and method of administration based on the formulation and availability. There is no guarantee that VIG will successfully treat of VIG therapy appears to be time dependent. VIG has not proven to be of benefit in the treatment of post-vaccinial encephalitis, and complications. At present, there are no other anti-viral therapies of proven benefit for the treatment of vaccinia-related complications.

# 4.2.2 Cidofovir (Vistide®, Gilead Sciences)

Cidofovir is an FDA-approved antiviral drug for the treatment of CMV retinitis among patients with AIDS. Cell-based in vitro studies and animal model studies have demonstrated this agent's antiviral activity against certain orthopoxviruses. Currently, its efficacy in the treatment of vaccinia-related complications in humans is unknown. According to the CDC, VIG is recommended as first line of therapy. Cidofovir may be considered as a secondary treatment, and will only be used when VIG therapy is not effective [Medical

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Management of Smallpox (Vaccinia) Vaccine Adverse Reactions: Vaccinia Immune Globulin and Cidofovir. Last updated September 28, 2009. Available at: <a href="http://www.bt.cdc.gov/agent/smallpox/vaccination/mgmt-adv-reactions.asp">http://www.bt.cdc.gov/agent/smallpox/vaccination/mgmt-adv-reactions.asp</a>]

## 5 BIOSPECIMEN COLLECTION

# 5.1 CORRELATIVE STUDIES FOR RESEARCH/PHARMACOKINETIC STUDIES

All patients enrolling will have blood samples drawn for PK studies and samples collected for the other studies as described below.

The plasma concentration-time data will be analyzed using WinNonlin software (Pharsight, Mountain View, CA). The maximum concentration, time to maximum concentration, the area under the curve extrapolated to infinity, and clearance will be calculated.

## 5.1.1 Collection of Specimens

before docetaxel administration, at approximately 5 minutes prior to the end of docetaxel infusion, and at 15 minutes, 30 minutes, 3h, One 6mL sodium heparin tube (BD, Franklin Lakes, NJ) is collected from each patient on Cycle 1 -at the following time points: 6h, 12h and 24h after the end of docetaxel infusion.

# 5.1.2 Handling and Processing of Specimen(s)

The samples will be placed immediately on wet ice and refrigerated. The date and exact time of each blood draw should be recorded on the sample tube and the PK sheet.

Please e-mail Julie Barnes at Julie.barnes@nih.gov and Paula Carter pcartera@mail.nih.gov at least 24 hours before transporting samples (the Friday before is preferred).

For sample pickup, page 102-11964.

For immediate help, call 240-760-6180 (main blood processing core number) or, if no answer, 240-760-6190 (main clinical pharmacology lab number).

For questions regarding sample processing, contact Julie Barnes by e-mail or at 240-760-6044.

Upon arrival in the Blood Processing Core, samples will be centrifuged, and the plasma transferred into cryovials for storage at -80C until the time of analysis. In addition, samples will be barcoded as described in section 5.3.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

The pharmacokinetic analysis will be performed on a research basis in the Blood Processing Core.

## 5.2 BIOMARKER STUDIES

5.2.1 Genetic Biomarkers

5.2.1.1 Collection of Specimens

One 6ml EDTA tube (BD, Franklin Lakes, NJ) will be collected from patients at baseline (after consent, prior to docetaxel or vaccinia initiation).

# 5.2.1.2 Handling and Processing of Specimens

Immediately after collection, invert the blood tube 8-10 times. Place the tube on wet ice and then store at 4°C in the refrigerator. The date and exact time of each blood draw should be recorded on the tube.

Please e-mail Julie Barnes at Julie. barnes@nih.gov and Paula Carter pcartera@mail.nih.gov at least 24 hours before transporting samples (the Friday before is preferred).

For sample pickup, page 102-11964.

For immediate help, call 240-760-6180 (main blood processing core number) or, if no answer, 240-760-6190 (main clinical pharmacology lab number).

For questions regarding sample processing, contact Julie Barnes by e-mail or at 240-760-6044.

Upon arrival in the BPC, genomic DNA will be extracted and analyzed for genetic polymorphisms.

The genotyping will be performed using DMET (Drug Metabolizing Enzymes and Transporters) array on a research basis in the Molecular Pharmacology Section.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## 5.2.2 Circulating Tumor Cells

# 5.2.2.1 Collection of Specimens for Veridex Analysis

CTC enumeration: Two 7cc lavender top tubes for flow-based CTC analysis will be collected before start of treatment (pre-docetaxel for Arm A, pre-vaccinia for Arm B & C), week 13 for Arm A & B, and week 9 for Arm C. Up to nine patients may have peripheral blood collected at the same time points in one 7.5cc CellSave Preservative Tube for Veridex CTC analysis.

# 5.2.2.2 Handling and Processing of Specimens for Veridex Analysis

trepel@helix.nih.gov; Min-Jung Lee at leemin@mail.nih.gov that the sample is scheduled. After the sample is drawn please call the Trepel lab at 240-760-6330 to communicate that the sample is ready. Keep the sample on the unit at room temperature. The sample CTC enumeration: As soon as possible after the patient is scheduled please send email notification to the Trepel lab: Jane Trepel at will be picked up by the lab and processed for CTC enumeration. The flow cytometric analyses will be performed by the Trepel laboratory. The Trepel lab will deliver CellSave tubes to the research nursing staff and arrange for sending the tubes for Veridex analysis.

# 5.2.2.3 Collection of Specimens for Epic Analysis

Arm C only: One 10ml Streck Cell-Free DNA (brown/black tube) will be collected from patients at baseline (pre-treatment), prior to docetaxel, and at completion of treatment.

# 5.2.2.3.1 Rationale of investigation for Epic Analysis

- Methods are in development for the purification and analysis of circulating tumor cells (CTC).
- slides, nucleated peripheral blood cells are attached to slides and examined, cytokeratin-positive/CD45-negative cells with an One of these novel CTC technologies, developed by Epic Sciences, is summarized as follows: whole blood is aliquoted onto recorded. This technology has the advantage of being able to identify cells that may be CTC but cytokeratin negative. Since intact nucleus and a malignancy-consistent morphology are identified as CTCs, and their exact positions on the slides positive or negative selection is not needed, all circulating cells are captured and analyzed via proprietary technology
- Multiplex analysis technologies have been developed to examine the levels and activities of androgen receptor.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

phenotype, such as AR splice variants, and how such changes are associated with clinical outcomes. The evaluation of CTCs may give valuable insight into how treatment affects changes in CTC

# 5.2.2.3.2 Handling and Processing of Specimens for Epic Analysis

PBMCs collected and stored at -80°C for immunology assays may also be shipped to Epic Sciences for CTC analysis. Samples will be The Blood Processing Core will be paged at 102-11964 for tube pick up and shipping via FedEx Priority Overnight to Epic Sciences. These samples will be sent in ambient shippers provided by Epic Sciences to keep samples at room temperature. Alternatively, shipped to the following address:

Epic Sciences Attn: Ryan Dittamore

9381 Judicial Drive, Ste. 200

San Diego, CA 92121

858-356-6610, ext. 124

## 5.2.3 Immunologic Parameters

- Antibodies to PSA, vaccinia, fowlpox may be tested
- Leukocyte CD3, CD4, CD8 subsets; CD4:CD8 ratio will be drawn at baseline and at each visit when on treatment and then at each follow-up visit while the patient remains on trial.
- Additional studies will include but are not limited to quantitative and qualitative assessments of regulatory T-cells, Natural Killers cells, Myeloid Derived Suppressor Cells, anti-glycan antibodies and Naïve T-cell/new thymic emigrants.
- Assessment of levels of cytokines.
- Immunologic studies will be repeated more frequently if clinically indicated, and any abnormalities potentially related to treatment will be followed until they have resolved, or have been determined not to be treatment-related.
- Peripheral blood mononuclear cells (PBMC):
- Intracellular cytokine staining assays for Brachyury-specific Tlymphocytes using PSA, MUC-1 and Brachyury-specific peptides CD3, CD4, CD8, and CD 19 subsets, NK markers and CD4:CD8 ratio.
- Phenotypic and functional analysis of immune cell subsets by flow cytometry.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## 5.2.3.1 Collection of Specimens

6 (10mL) green top sodium heparin tubes for PBMC; 2 (8mL) SST tubes for serum sample will be collected as follows:

- Arm A
- o Baseline (pre-treatment), post 3 and 6 cycles of docetaxel (week 10 and 19), post 1st dose of PROSTVAC-F (week 24), at completion of treatment, and every 6 months until progression.
- Arm B:
- o Baseline (pre-treatment), post 1<sup>st</sup> dose of PROSTVAC-F (week 4), at completion of treatment (week 19), and every 6 months until progression.
- Arm C
- Baseline (pre-treatment), post 1st dose of PROSTVAC-F (week 6), pre-docetaxel, post 3 cycles of docetaxel (chemo week 10), at completion of treatment, and every 6 months until progression.

# 5.2.3.2 Handling and Processing of Specimen(s)

The samples will be processed through:

Clinical Services Program

NCI Frederick Cancer Research and Development Center

PO Box B

Frederick, MD 21702

301-846-1000

On days samples are drawn, Jen Bangh at CSP should be notified (phone: [301] 846-5893; fax [301] 846-6222). She will arrange same-day courier delivery of the specimens. The research samples will contain labels on the blood tubes that have the patient's initials, date of birth, the assigned protocol, and the date the sample was drawn. The transmittal forms accompanying the samples also contain the same information.

Once a patient's treatment schedule has been determined, it should be faxed to Caroline Jochems at the Laboratory of Tumor Immunology and Biology/ NIH (Fax: [301] 496-2756; phone: [301] 496-9573) for planning purposes.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## 5.2.3.3 Immunologic Assays

## 5.2.3.3.1 Sera Antibody Analysis:

Serum will be stored at -80 degrees Celsius and there will be planned analysis for generation of antibodies to PSA, BCG, PAP, PSMA, PSCA, and/or MUC-1.

## 5.2.3.4 Natural Killer (NK) CELLS

The number and phenotype of NK cells will be determined by phenotypic analysis of PMBCs stained for CD56, CD3, CD8, and CD16 by flow cytometry.

### 5.2.3.5 Immune Subsets

Subsets of immune cells will also be followed in response to treatment.

## 5.2.3.6 Regulatory T Cells

responses. Higher levels of regulatory T-cells have been reported in the peripheral blood mononuclear cells of patients with several types of tumors. The number and phenotype of regulatory T-cells in peripheral blood mononuclear cells from patients in this study containing 3% fetal bovine serum) and stained for CD4, CD25, CD127, FoxP3, CTLA-4, CD45RA, and CD8. The ratios between regulatory T-cells and CD4 effector cells and the ratios between regulatory T-cells and CD8 Effector cells will also be analyzed. will be determined by 7-color flow cytometry analysis. Cells will be resuspended in staining buffer (phosphate-buffered saline Regulatory T cells have been shown to inhibit the activation and function of T cells that participate in antigen-specific immune

### 5.2.3.7 Additional Assays

analysis of immune-cell subsets and analyses for cytokines (IFN-γ, IL-10, IL-12, IL-2, IL-4, etc.), chemokines, antibodies related to Blood samples may be used for additional research studies, which may include one of the following - phenotypic and functional the tumor or vaccine, tumor associated antigens related to the tumor or the vaccine, and/or other immune response markers.

### 5.2.3.8 Biopsy Analysis

will assess immune responses in the tumor microenvironment using immune histochemistry as the primary analysis and could include When logistically feasible, consenting patients will have a biopsy prior to treatments and after 2 months of vaccine. Biopsy findings

Biopsy sites will vary based on patient and the location of disease. Sites could include intraprostatic tumors or metastatic sites. Biopsies will be limited to 1 site (although a biopsy within the prostate itself may have up to 3 or 4 lesions to be biopsied)

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## 5.2.3.8.1 Immunohistochemistry

The Laboratory of Pathology and the Warren G. Magnuson Clinical Center will perform Immunohistochemistry on biopsied tissue, if the patient elects to have the procedure. Immunohistochemistry of these tissue specimens will be obtained for CD4, CD8, and FOX-P3. In addition, phenotypic analysis of infiltrating immune cells will be performed.

Immunohistologic grading schema of the lesions

| Score | %positive cells of each subtyp |
|-------|--------------------------------|
| 0 | 0 |
| _ | 1-25% |
| 2 | 26-50% |
| c | >50% |

All staining will be categorized as being membrane or nuclear

# .3 SAMPLE STORAGE, TRACKING AND DISPOSITION

available, the CRIS downtime procedures will be followed. Samples will not be sent outside NIH without IRB notification and an Samples will be ordered in CRIS and tracked through the Clinical Trial Data Management System. Should a CRIS screen not be executed MTA.

## 5.3.1 Blood Processing Core - Storage

LabSamples) utilized by the BPC. This is a secure program, with access to LABrador limited to defined Figg lab personnel, who are issued individual user accounts. Installation of LABrador is limited to computers specified by Dr. Figg. These computers all have a password restricted login screen. All Figg lab personnel with access to patient information annually complete the NIH online All samples sent to the Blood Processing Core (BPC) will be barcoded, with data entered and stored in the LABrador (aka Protection of Human Subjects course. LABrador creates a unique barcode ID for every sample and sample box, which cannot be traced back to patients without LABrador access. The data recorded for each sample includes the patient ID, name, trial name/protocol number, time drawn, cycle time point, dose, material type, as well as box and freezer location. Patient demographics associated with the clinical center patient number are

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

provided in the system. For each sample, there are notes associated with the processing method (delay in sample processing, storage conditions on the ward, etc.)

Barcoded samples are stored in barcoded boxes in a locked freezer at either -20 or -80°C according to stability requirements. These freezers are located onsite in the BPC and offsite at NCI Frederick Central Repository Services in Frederick, MD. Visitors to the laboratory are required to be accompanied by laboratory staff at all times.

used for research purposes associated with this trial (as per the IRB approved protocol) and that any unused samples must be returned to the BPC. It is the responsibility of the NCI Principal Investigator to ensure that the samples requested are being used in a manner requests are monitored and tracked in LABrador. All researchers are required to sign a form stating that the samples are only to be Access to stored clinical samples is restricted. Samples will be stored until requested by a researcher named on the protocol. All consistent with IRB approval.

Following completion of this study, samples will remain in storage as detailed above. Access to these samples will only be granted following IRB approval of an additional protocol, granting the rights to use the material.

provide a written request. Following receipt of this request, the samples will be destroyed (or returned to the patient, if so requested), and reported as such to the IRB. Any samples lost (in transit or by a researcher) or destroyed due to unknown sample integrity (i.e. If, at any time, a patient withdraws from the study and does not wish for their existing samples to be utilized, the individual must broken freezer allows for extensive sample thawing, etc.) will be reported as such to the IRB.

Sample barcodes are linked to patient demographics and limited clinical information. This information will only be provided to information such as race, age, dates of diagnosis and death, and histological information about the tumor, in order to correlate investigators listed on this protocol, via registered use of the LABrador. It is critical that the sample remains linked to patient genotype with these variables.

# 5.3.2 Handling and Storage for Research Samples Managed by Jane Trepel's Laboratory

Using a secure laboratory computerized database and a backup hardcopy process, all specimen collection and processing steps are documented and the specific location of each specimen is tracked. Each new specimen collected is assigned a unique 2D barcode identifier that can be linked to the original specimen collected and other relevant information within the inventory system. To ensure patient confidentiality, only containers used for the initial specimen collections will be labeled with patient identifiers. De-identified labels will be applied to all subsequent specimen containers. When specimens are processed and aliquoted, no patient information will be included on the new containers. Original specimen containers will be discarded. Only de-linked specimens will be stored. The inventory process contains other security provisions sufficient to safeguard patient privacy and confidentiality. Access to the

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

inventory system and associated documents is restricted to appropriate personnel only. SOPs ensure that any changes in the informed consent made by a patient and relayed to the PI will be reflected in the inventory system to ensure that specimens are destroyed as appropriate. All laboratory personnel are trained to adhere to SOPs and are monitored for high-quality performance.

# 5.3.3 Samples Sent to Clinical Services Program (CSP)

All data associated with patient samples are protected by a secure database. All samples drawn at the NIH Clinical Center will be transported to the NCI Frederick Central Repository by Leidos couriers. Samples will be tracked and managed by the Central Repository database. All samples will be stored in liquid nitrogen. These freezers are located at NCI Frederick Central Repository in Frederick, Maryland.

American Type Culture Collection (ATCC) manages the NCI-Frederick Central Repositories under subcontract to Leidos Biomedical Research, Inc. NCI-Frederick Central Repositories store, among other things, biological specimens in support of NIH clinical studies. All specimens are stored in secure, limited access facilities with sufficient security, back up and emergency support capability and monitoring to ensure long-term integrity of the specimens for research. ATCC role is limited to clinical research databases and repositories containing patient specimens. ATCC does not conduct nor has any vested interest in research on human subjects, but does provide services and support the efforts of its customers, many of which are involved in research on human subjects.

It is the intent and purpose of ATCC to accept only de-identified samples and sample information. To the limit of our ability, every effort will be made to ensure that protected information is not sent electronically or by hard copy or on vial labels. Sample data is stored in the BioSpecimen Inventory System II (BSI). This inventory tracking system is used to manage the storage and specimens received by the repository. If a specimen goes out of the inventory, the system maintains data associated with the withdraw multi-user environment for tracking millions of specimens. The system controls how and in what order database updates and searches tracking for processes that are done to specimens including shipping, returning to inventory, aliquoting, thawing, additives, and other access levels, and 36 user permissions (levels of access) that can be set to control access to the system functions. BSI provides audit are performed. This control prevents deadlocks and race conditions. For security, BSI has user password access, three types of user retrieval of specimens as well as maintain specimen data. BSI is designed for controlled, concurrent access. It provides a real-time, processes. BSI tracks the ancestry of specimens as they are aliquoted, as well as discrepancies and discrepancy resolution for

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

request. Vials are labeled with a unique BSI ID which is printed in both eye readable and bar coded format. No patient specific information is encoded in this ID.

specimens for which they have not been authorized. Access to specimen storage is confined to repository staff. Visitors to the Investigators are granted view, input and withdraw authority only for their specimens. They may not view specimen data or access repositories are escorted by repository staff at all times.

# 5.3.4 Protocol Completion/Sample Destruction

Once primary research objectives for the protocol are achieved, intramural researchers can request access to remaining samples, provided they have an IRB-approved protocol and patient consent.

consent. Samples will also be reported as lost if they are lost in transit or misplaced by a researcher. Freezer problems, lost samples or participant's data will be excluded from future distributions, but data that have already been distributed for approved research use will other problems associated with samples will also be reported to the IRB, the NCI Clinical Director, and the office of the CCR, NCI. Samples and associated data will be stored permanently unless the patient withdraws consent. If the patient withdraws consent the environmental conditions (ex. broken freezer or lack of dry ice in shipping container) or if a patient chooses to withdraw his/her not be able to be retrieved. The PI will report destroyed samples to the IRB if samples become unsalvageable or destroyed by

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# DATA COLLECTION AND EVALUATION

### .1 DATA COLLECTION

- Eligible patients must be confirmed and checklist completed. Consent form must be signed prior to registration with Central Registration Office.
- Data will be secured in NCI C3D database. Data will be collected using protocol-specific case report forms, and verified for secured electronic data base. The following protocol-specific study forms will be complete and stored: eligibility checklist accuracy and completeness. Hard copies of data will be stored in locked secured areas and data will be entered onto a (developed by Central Registration Office, CRO). A copy of all serious AE forms will be kept in the research record. 6.1.2
- Treatment is given according to protocol (dated notes about doses given, complications, and clinical outcomes).
- 5.1.4 Toxicity is assessed according to protocol (laboratory report slips, etc.)
- Response is assessed according to protocol (X-ray, scan, lab reports, and date noted on clinical assessment, as appropriate).
- i.1.6 Drug Accountability Records are kept for each patient.
- For Arm A patients, who have not yet received PROSTVAC, we will only collect adverse events that are serious and/or unexpected. Once patients begin the PROSTVAC injection, adverse events will be collected as outlined in Section 7. 6.1.7

The PI will be responsible for overseeing entry of data into an in-house password protected electronic system (C3D) and ensuring data network drives or in approved alternative sites that comply with NIH security standards. Primary and final analyzed data will have manager will assist with the data management efforts. All data obtained during the conduct of the protocol will be kept in secure accuracy, consistency and timeliness. The principal investigator, associate investigators/research nurses and/or a contracted data identifiers so that research data can be attributed to an individual human subject participant.

followed until return to baseline or stabilization of event. Patients will be followed for adverse events for 30 days after removal from All adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity, will be study treatment or until off-study, whichever comes first. End of study procedures: Data will be stored according to HHS, FDA regulations, and NIH Intramural Records Retention Schedule

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Loss or destruction of data: Should we become aware that a major breach in our plan to protect subject confidentiality and trial data has occurred, the IRB will be notified

## 6.2 DATA SHARING PLANS

6.2.1 Human Data Sharing Plan

### What data will be shared?

I will share human data generated in this research for future research as follows:

 $\boxtimes$  De-identified data in an NIH-funded or approved public repository.

□ De-Identified data in BTRIS (automatic for activities in the Clinical Center)

## How and where will the data be shared?

Data will be shared through

National problem of Publications Section 2.

## When will the data be shared?

⊠ Before publication.

 $\boxtimes$  At the time of publication or shortly thereafter.

### 3 RESPONSE CRITERIA

Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [31] and Prostate Cancer Clinical Trials Working Group criteria Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

(PCWG2) [32]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

#### 6.3.1 Definitions

Evaluable for toxicity: All patients will be evaluable for toxicity from the time of their first treatment

response classified according to the definitions stated below. (Note: Patients who exhibit objective disease progression prior to the cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. These patients will have their Evaluable for objective response: Only those patients who have measurable disease present at baseline, have received at least one end of cycle 1 will also be considered evaluable.)

considered evaluable for non-target disease. The response assessment is based on the presence, absence, or unequivocal progression Evaluable Non-Target Disease Response: Patients who have lesions present at baseline that are evaluable but do not meet the definitions of measurable disease, have received at least one cycle of therapy, and have had their disease re-evaluated will be of the lesions.

### 6.3.2 Disease Parameters

Measurable disease: Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded:

- By chest x-ray:  $\geq 20$  mm;
- By CT scan:
- o Scan slice thickness 5 mm or under: as  $\geq 10$  mm
- Scan slice thickness >5 mm: double the slice thickness
- With calipers on clinical exam:  $\geq 10 \text{ mm}$ .

All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

<u>Malignant lymph nodes.</u> To be considered pathologically enlarged and measurable, a lymph node must be  $\geq 15$  mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

pleural/pericardial effusions, lymphangitis cutis/pulmonitis, inflammatory breast disease, and abdominal masses (not followed by CT lymph nodes with  $\geq 10$  to <15 mm short axis), are considered non-measurable disease. Bone lesions, leptomeningeal disease, ascites, Non-measurable disease. All other lesions (or sites of disease), including small lesions (longest diameter <10 mm or pathological or MRI), are considered as non-measurable.

Note: Cystic lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.

measurability described above. However, if non-cystic lesions are present in the same patient, these are preferred for selection as 'Cystic lesions' thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of target lesions.

baseline sum diameters will be used as reference to further characterize any objective tumor regression in the measurable dimension of organs, should be identified as target lesions and recorded and measured at baseline. Target lesions should be selected on the basis of sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported Target lesions. All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved reproducible measurement in which circumstance the next largest lesion which can be measured reproducibly should be selected. as the baseline sum diameters. If lymph nodes are to be included in the sum, then only the short axis is added into the sum. The themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to their size (lesions with the longest diameter), be representative of all involved organs, but in addition should be those that lend

Non-target lesions. All other lesions (or sites of disease) including any measurable lesions over and above the 5 target lesions should be identified as **non-target lesions** and should also be recorded at baseline. Measurements of these lesions are not required, but the presence, absence, or in rare cases unequivocal progression of each should be noted throughout follow-up.

# 6.3.3 Methods for Evaluation of Measurable Disease

performed as closely as possible to the beginning of treatment and never more than 8 weeks before the beginning of the treatment. All measurements should be taken and recorded in metric notation using a ruler or calipers. All baseline evaluations should be

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination unless the lesion(s) being followed The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline cannot be imaged but are assessable by clinical exam. Clinical lesions: Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes) and ≥10 mm diameter as assessed using calipers (e.g., skin nodules). In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.

Chest x-ray: Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT is preferable.

thickness is 5 mm or less. If CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be Conventional CT and MRI: This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice twice the slice thickness. MRI is also acceptable in certain situations (e.g. for body scans).

should be the same as was used at baseline and the lesions should be measured/assessed on the same pulse sequence. It is beyond the Ideally, the same type of scanner should be used and the image acquisition protocol should be followed as closely as possible to prior used should be optimized for the evaluation of the type and site of disease. Furthermore, as with CT, the modality used at follow-up availability of MRI is variable globally. As with CT, if an MRI is performed, the technical specifications of the scanning sequences acquisition variables involved in MRI, which greatly impact image quality, lesion conspicuity, and measurement. Furthermore, the Use of MRI remains a complex issue. MRI has excellent contrast, spatial, and temporal resolution; however, there are many image scope of the RECIST guidelines to prescribe specific MRI pulse sequence parameters for all scanners, body parts, and diseases. scans. Body scans should be performed with breath-hold scanning techniques, if possible. <u>PET-CT:</u> At present, the low dose or attenuation correction CT portion of a combined PET-CT is not always of optimal diagnostic CT identical diagnostic quality to a diagnostic CT (with IV and oral contrast), then the CT portion of the PET-CT can be used for RECIST quality for use with RECIST measurements. However, if the site can document that the CT performed as part of a PET-CT is of however, that the PET portion of the CT introduces additional data which may bias an investigator if it is not routinely or serially measurements and can be used interchangeably with conventional CT in accurately measuring cancer lesions over time. Note

identified by ultrasound in the course of the study, confirmation by CT or MRI is advised. If there is concern about radiation exposure examinations cannot be reproduced in their entirety for independent review at a later date and, because they are operator dependent, it Ultrasound: Ultrasound is not useful in assessment of lesion size and should not be used as a method of measurement. Ultrasound cannot be guaranteed that the same technique and measurements will be taken from one assessment to the next. If new lesions are at CT, MRI may be used instead of CT in selected instances.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

techniques may be useful to confirm complete pathological response when biopsies are obtained or to determine relapse in trials where Endoscopy, Laparoscopy: The utilization of these techniques for objective tumor evaluation is not advised. However, such recurrence following complete response (CR) or surgical resection is an endpoint.

recurrent ovarian cancer) and PSA response (in recurrent prostate cancer) have been published [32-34]. In addition, the Gynecologic <u>Tumor markers:</u> Tumor markers alone cannot be used to assess response. If markers are initially above the upper normal limit, they Cancer Intergroup has developed CA-125 progression criteria which are to be integrated with objective tumor assessment for use in must normalize for a patient to be considered in complete clinical response. Specific guidelines for both CA-125 response (in first-line trials in ovarian cancer [35].

Cytology, Histology: These techniques can be used to differentiate between partial responses (PR) and complete responses (CR) in rare cases (e.g., residual lesions in tumor types, such as germ cell tumors, where known residual benign tumors can remain)

tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease (an effusion may The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable be a side effect of the treatment) and progressive disease.

PET scanning to complement CT scanning in assessment of progression (particularly possible 'new' disease). New lesions on the basis FDG-PET: While FDG-PET response assessments need additional study, it is sometimes reasonable to incorporate the use of FDGof FDG-PET imaging can be identified according to the following algorithm:

- Negative FDG-PET at baseline, with a positive FDG-PET at follow-up is a sign of PD based on a new lesion.
- disease on CT, additional follow-up CT scans are needed to determine if there is truly progression occurring at that site (if new site of disease confirmed by CT, this is PD. If the positive FDG-PET at follow-up is not confirmed as a new site of corresponds to a pre-existing site of disease on CT that is not progressing on the basis of the anatomic images, this is not No FDG-PET at baseline and a positive FDG-PET at follow-up: If the positive FDG-PET at follow-up corresponds to a so, the date of PD will be the date of the initial abnormal FDG-PET scan). If the positive FDG-PET at follow-up
- prospectively described in the protocol and supported by disease-specific medical literature for the indication. However, it radiographic abnormality is thought to represent fibrosis or scarring. The use of FDG-PET in this circumstance should be must be acknowledged that both approaches may lead to false positive CR due to limitations of FDG-PET and biopsy FDG-PET may be used to upgrade a response to a CR in a manner similar to a biopsy in cases where a residual resolution/sensitivity. ပ

Note: A 'positive' FDG-PET scan lesion means one which is FDG avid with an uptake greater than twice that of the surrounding tissue on the attenuation corrected image.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

### 6.3.4 Response Criteria

## 6.3.4.1 Evaluation of Target Lesions

Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of

on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also <u>Progressive Disease (PD)</u>: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions)

Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.

## 6.3.4.2 Evaluation of Non-Target Lesions

Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).

Note: If tumor markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response. Non-CR/Non-PD: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.

Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. not a single lesion increase. Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or Principal Investigator)

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## 6.3.4.3 Metastatic Bone Lesions

declaring disease progression by bone scan. 36 Confirmatory scans may not be necessary in the presence of progressive soft tissue disease or the appearance of multiple new bone lesions that in the opinion of the investigator are consistent with a progressive overall clinical course. bone scan and controlling for tumor flare. 36 PCWG2 defines disease progression as the appearance of two or more lesions on bone scan. "tumor flare" phenomenon. Thus, PCWG2 recommends that a repeat scan performed 6 or more weeks later should be performed before The Prostate Cancer Working Group 2 (PCWG2) criteria published guidelines on measuring treatment effects on bone metastases using However, new lesions seen on the first post-treatment bone scan may represent disease that was not detected on the pre-study scan or a

For this study, if a patient has new lesions on the first post-treatment bone scan, they may remain on-study with the first post-treatment bone clinically indicated and compared to the new baseline (first post-treatment scan) in determining disease progression by bone scan. Should the subsequent scans show 2 or more new lesions relative to the new baseline, the patient will then meet progression criteria. The date of scan now becoming the new baseline for future evaluations. All subsequent scans can be conducted as scheduled in the protocol or as disease progression is recorded as the date of the first scan when the new lesions are first detected.36

# 6.3.4.4 Evaluation of Best Overall Response

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

# For Patients with Measurable Disease (i.e., Target Disease)

| Target<br>Lesions | Non-Target<br>Lesions | New<br>Lesions | New Overall Lesions Response | Best Overall Response when<br>Confirmation is Required* |
|---|---|---|---|---|
| CR | CR | No | CR | ≥4 wks. Confirmation** |
| CR | Non-<br>CR/Non-PD | No | PR | |
| CR | Not<br>evaluated | No | PR | ≥4 wks. Confirmation** |
| PR | Non-<br>CR/Non- | No | PR | |


| | Documented at least once >4 wks. from baseline** | | no prior SD, PR or CR | | See RECIST 1.1 manuscript for further details on what is evidence of a new lesion. | Only for non-randomized trials with response as primary endpoint. | In exceptional circumstances, unequivocal progression in non-target lesions may be accepted as disease progression. | Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment. |
|---|---|---|---|---|---|---|---|---|
| | SD | PD | PD | PD | for further d | ıls with resp | , unequivoca<br>isease progra | ration of hes<br>without obje<br>Id be reporte<br>should be m |
| | No | Yes or<br>No | Yes or<br>No | Yes | anuscript | omized tria | umstances,<br>epted as di | bal deterio<br>treatment v<br>time shoul<br>very effort<br>fter discon |
| PD/not<br>evaluated | Non-<br>CR/Non-<br>PD/not<br>evaluated | Any | PD*** | Any | See RECIST 1.1 m<br>new lesion. | ıly for non-rando | In exceptional circumstances, unequivocal proglesions may be accepted as disease progression. | Patients with a global deterioration of health status is discontinuation of treatment without objective evide progression at that time should be reported as "symp deterioration." Every effort should be made to doe progression even after discontinuation of treatment. |
| | SD | PD | Any | Any | * See | ** On | *** In e | Note: Pat dis dis det det pro |

# For Patients with Non-Measurable Disease (i.e., Non-Target Disease)

| Overall Response |
|--------------------|
| New Lesions |
| Non-Target Lesions |


| CR | No | CR |
|-------------------|-----------|----------------|
| Non-CR/non-PD | No | Non-CR/non-PD* |
| Not all evaluated | No | not evaluated |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

since SD is increasingly used as an endpoint for assessment of efficacy in some trials so to assign this category when no lesions can be measured is not advised \* 'Non-CR/non-PD' is preferred over 'stable disease' for non-target disease

## 6.3.5 Duration of Response

(whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for Duration of overall response: The duration of overall response is measured from the time measurement criteria are met for CR or PR progressive disease the smallest measurements recorded since the treatment started)

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented. Duration of stable disease: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.

## 6.3.6 Serologic Response:

PSA will be assessed at each visit during treatment and every 12 weeks thereafter. Patients will be assigned response based on the following criteria.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Complete Serological Response: PSA level less than 0.2 ng/ml measured for 2 consecutive measurements at least 4 weeks apart.

Serological Partial Response: decline of PSA at least 50% measured for 2 consecutive measurements at least 4 weeks apart.

Serological Progression:

- PSA has risen above 4 ng/ml or an increase in PSA of more than 50% above nadir (lowest PSA on ADT) or confirmed rise in PSA.
- Values must be measured for 2 consecutive measurements at least 2 weeks apart.
- The date of the first increase will be recorded as progression.

Time to Serologic Progression will be defined as interval between initiation of ADT and date of PSA progression or death from any

### 6.4 TOXICITY CRITERIA

will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 The following adverse event management guidelines are intended to ensure the safety of each patient while on the study. The (http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc\_40) the CTCAE version 4.0 can be downloaded from the CTEP web site

## 6.5 ANTIGEN SPREAD SCORING

As described in section 1.2.5 of the background, antigen spread will be evaluated using CD4 and CD8 analysis of CD107a expression specifically by the vaccine (MUC1 and Brachyury) they will be weighted 150% of the PSA responses. The scoring parameters are and IFN- $\gamma$ , IL-2 and TNF- $\alpha$  intracellular cytokine staining. In order to give added weight to the spread antigens not targeted below with a possible maximum score of 30.

#### For PSA:

1 point each of the four CD4 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 4

1 point each of the four CD8 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 4

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Total possible score for PSA response is 8

#### For MUC1:

1.5 points each of the four CD4 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 6

1.5 points each of the four CD8 parameters (CD107a, IFN-γ, IL-2 and TNF-α) – max total of 6

Total possible score for PSA response is 12.

#### For Brachyury:

1.5 points each of the four CD4 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 6

1.5 points each of the four CD8 parameters (CD107a, IFN- $\gamma$ , IL-2 and TNF- $\alpha$ ) – max total of 6

Total possible score for PSA response is 12.

# SAFETY REPORTING REQUIREMENTS/DATA AND SAFETY MONITORING PLAN

#### .1 DEFINITIONS

#### 7.1.1 Adverse Event

laboratory finding), symptom, or disease, temporally associated with the subject's participation in research, whether or not considered Any untoward medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or related to the subject's participation in the research.

## 7.1.2 Suspected adverse reaction

For the purposes of IND safety reporting, 'reasonable possibility' means there is evidence to suggest a causal relationship between the Suspected adverse reaction means any adverse event for which there is a reasonable possibility that the drug caused the adverse event. drug and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

## 7.1.3 Unexpected adverse reaction

An adverse event or suspected adverse reaction is considered "unexpected" if it is not listed in the investigator brochure or is not listed adverse events or suspected adverse reactions that are mentioned in the investigator brochure as occurring with a class of drugs or as the risk information described in the general investigational plan or elsewhere in the current application. "Unexpected" also refers to at the specificity or severity that has been observed; or, if an investigator brochure is not required or available, is not consistent with anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation.

#### 7.1.4 Serious

An Unanticipated Problem or Protocol Deviation is serious if it meets the definition of a Serious Adverse Event or if it compromises the safety, welfare or rights of subjects or others.

## 7.1.5 Serious Adverse Event

An adverse event or suspected adverse reaction is considered serious if in the view of the investigator or the sponsor, it results in any of the following:

- Death,
- A life-threatening adverse drug experience
- Inpatient hospitalization or prolongation of existing hospitalization
- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- A congenital anomaly/birth defect.
- serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the patient or subject Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 7.1.6 Disability

A substantial disruption of a person's ability to conduct normal life functions.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 7.1.7 Life-threatening adverse drug experience

immediate risk of death from the reaction as it occurred, i.e., it does not include a reaction that had it occurred in a more severe form, Any adverse event or suspected adverse reaction that places the patient or subject, in the view of the investigator or sponsor, at might have caused death.

## 7.1.8 Protocol Deviation (NIH Definition)

Any change, divergence, or departure from the IRB-approved research protocol.

## 7.1.9 Non-compliance (NIH Definition)

The failure to comply with applicable NIH Human Research Protections Program (HRPP) policies, IRB requirements, or regulatory requirements for the protection of human research subjects.

## 7.1.10 Unanticipated Problem

Any incident, experience, or outcome that:

- Is unexpected in terms of nature, severity, or frequency in relation to
- (a) the research risks that are described in the IRB-approved research protocol and informed consent document; Investigator's Brochure or other study documents, and
- (b) the characteristics of the subject population being studied; AND
- Is related or possibly related to participation in the research; AND
- Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

# .2 NIH-IRB AND CLINICAL DIRECTOR (CD) REPORTING

7.2.1 NIH-IRB and NCI CD Expedited Reporting of Unanticipated Problems and Deaths

The Protocol PI will report in the NIH Problem Form to the NIH-IRB and NCI CD:

- All deaths, except deaths due to progressive disease
- All Protocol Deviations

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- All Unanticipated Problems
- All non-compliance

Reports must be received within 7 days of PI awareness via iRIS.

7.2.2 NIH-IRB Requirements for PI Reporting at Continuing Review

The protocol PI will report to the NIH-IRB:

- A summary of all protocol deviations in a tabular format to include the date the deviation occurred, a brief description of the deviation and any corrective action.
- 2. A summary of any instances of non-compliance
- 3. A tabular summary of the following adverse events:
- All Grade 2 unexpected events that are possibly, probably or definitely related to the research;
- All Grade 3 and 4 events that are possibly, probably or definitely related to the research;
- All Grade 5 events regardless of attribution;
- All Serious Events regardless of attribution.

NOTE: Grade 1 events are not required to be reported.

# 7.2.3 NIH-IRB Reporting of IND Safety Reports

Only IND Safety Reports that meet the definition of an unanticipated problem will need to be reported to the NIH IRB.

# 7.3 IND SPONSOR REPORTING CRITERIA

sponsor, using the mandatory MedWatch form 3500a or equivalent, any serious adverse event, whether or not considered drug related, During the first 30 days after the subject receives investigational agent/intervention, the investigator must immediately report to the possibility that the drug caused the event. For serious adverse events that occur more than 30 days after the last administration of investigational agent/intervention, only report those that have an attribution of at least possibly related to the agent/intervention. including those listed in the protocol or investigator brochure and must include an assessment of whether there is a reasonable

Required timing for reporting per the above guideline:

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Deaths (except death due to progressive disease) must be reported via email within 24 hours. A complete report must be submitted within one business day.

Other serious adverse events as well as deaths due to progressive disease must be reported within one business day

Study endpoints that are serious adverse events (e.g. all-cause mortality) must be reported in accordance with the protocol unless there is evidence suggesting a causal relationship between the drug and the event (e.g. death from anaphylaxis). In that case, the investigator must immediately report the death to the sponsor.

Events will be submitted to the Center for Cancer Research (CCR) at: CCRsafety@mail.nih.gov and to the CCR PI and study coordinator.

7.3.1 Reporting Pregnancy

7.3.1.1 Paternal exposure

Male patients should refrain from fathering a child or donating sperm during the study and for 4 months after the last dose of (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth, or congenital abnormality) occurring from the date of PROSTVAC. Pregnancy of the patient's partner is not considered to be an AE. However, the outcome of all pregnancies the first dose until 4 months after the last dose should, if possible, be followed up and documented.

## SAFETY REPORTING CRITERIA TO THE PHARMACEUTICAL COLLABORATORS 7.4

All events listed below must be reported in the defined timelines to CCRsafety@mail.nih.gov.

The CCR Office of Regulatory Affairs will send all reports to the manufacturer as described below.

1.1.1 Reporting to Bavarian Nordic, Inc.

The investigator should submit all safety reports that are sent to the FDA using the Medwatch 3500 Form to:

Bavarian Nordic, Inc.

Email: pharmacovigilance@bavarian-nordic.com;

Fax number for pharmacovigilance at BN: 888-465-1219

Attention: Karen Latina

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 5 INSTITUTIONAL BIOSAFETY COMMITTEE (IBC) REPORTING CRITERIA

# .5.1 Serious Adverse Event Reports to IBC

events that are unexpected and associated with the use of the PROSTVAC, but are not fatal or life-threatening, must be reported to the The Principal Investigator (or delegate) will notify IBC of any unexpected fatal or life-threatening experience associated with the use NIH IBC as soon as possible, but not later than 15 calendar days after the investigator's initial receipt of the information. Adverse of PROSTVAC as soon as possible but in no event later than 7 calendar days of initial receipt of the information. Serious adverse events may be reported by using the FDA Form 3500a.

## 7.5.2 Annual Reports to IBC

Alternatively, the IRB Continuing Review report can be sent to the IBC in lieu of a separate report. Please include the IBC protocol Within 60 days after the one-year anniversary of the date on which the IBC approved the initial protocol, and after each subsequent anniversary until the trial is completed, the Principal Investigator (or delegate) shall submit the information described below. number on the report.

## 7.5.2.1 Clinical Trial Information

A brief summary of the status of the trial in progress or completed during the previous year. The summary is required to include the following information:

- the title and purpose of the trial
- clinical site
- the Principal Investigator
- clinical protocol identifiers
- participant population (such as disease indication and general age group, e.g., adult or pediatric);
- the total number of participants planned for inclusion in the trial; the number entered into the trial to date whose participation in the trial was completed; and the number who dropped out of the trial with a brief description of the reasons
- the status of the trial, e.g., open to accrual of subjects, closed but data collection ongoing, or fully completed,
- if the trial has been completed, a brief description of any study results.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 7.5.2.2 Progress Report and Data Analysis

Information obtained during the previous year's clinical and non-clinical investigations, including:

- a narrative or tabular summary showing the most frequent and most serious adverse experiences by body system
- a summary of all serious adverse events submitted during the past year
- a summary of serious adverse events that were expected or considered to have causes not associated with the use of the gene transfer product such as disease progression or concurrent medications
- if any deaths have occurred, the number of participants who died during participation in the investigation and causes of death
  - a brief description of any information obtained that is pertinent to an understanding of the gene transfer product's actions, including, for example, information about dose-response, information from controlled trials, and information about

# 6 DATA AND SAFETY MONITORING PLAN

# 7.6.1 Principal Investigator/Research Team

patient. Decisions about dose level enrollment and dose escalation if applicable will be made based on the toxicity data from prior The clinical research team will meet on a regular basis weekly when patients are being actively treated on the trial to discuss each

events will be reported as required above. Any safety concerns, new information that might affect either the ethical and or scientific All data will be collected in a timely manner and reviewed by the principal investigator or a lead associate investigator. Adverse conduct of the trial, or protocol deviations will be immediately reported to the IRB using iRIS.

principal investigator will personally conduct or supervise the investigation and provide appropriate delegation of responsibilities to The principal investigator will review adverse event and response data on each patient to ensure safety and data accuracy. The other members of the research staff.

## 7.6.2 Sponsor Monitoring Plan

confirmation of: study data, specifically data that could affect the interpretation of primary study endpoints; adherence to the protocol, As a sponsor for clinical trials, FDA regulations require the CCR to maintain a monitoring program. The CCR's program allows for

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

regulations, and SOPs; and human subjects protection. This is done through independent verification of study data with source documentation focusing on:

- Informed consent process
- Eligibility confirmation
- Drug administration and accountability
- Adverse events monitoring
- Response assessment.

The monitoring program also extends to multi-site research when the CCR is the coordinating center.

This trial will be monitored by personnel employed by an NCI contractor. Monitors are qualified by training and experience to monitor the progress of clinical trials. Personnel monitoring this study will not be affiliated in any way with the trial conduct.

# 7.6.3 Safety Monitoring Committee (SMC)

This protocol will require oversight from the Safety Monitoring Committee (SMC). Initial review will occur as soon as possible after meeting schedule permits or more frequently as may be required by the SMC. For initial and subsequent reviews, protocols will not be reviewed if there is no accrual within the review period. Written outcome letters will be generated in response to the monitoring the annual NIH-IRB continuing review date. Subsequently, each protocol will be reviewed as close to annually as the quarterly activities and submitted to the Principal investigator and Clinical Director or Deputy Clinical Director, CCR, NCI

# STATISTICAL CONSIDERATIONS

#### 8.1 ARMS A AND B

considered positive (from 0 to 30 as described in section 1.2.5 and 6.5), and called the response score, determined for each patient at The primary objective of this trial is to determine if PROSTVAC when combined with docetaxel can induce antigen spreading or a much greater response than docetaxel alone; thus, the objective will be to determine if a large difference in results may be observed 19 weeks following treatment initiation. It is anticipated that combining PROSTVAC with docetaxel (combination) may induce a docetaxel then PROSTVAC. The main endpoint will be the mean over all patients, by arm, of the sum of the individual antigens randomized to either ADT followed by simultaneous docetaxel + PROSTVAC (combination) or ADT followed by sequential greater breadth of immune response compared to docetaxel followed by PROSTVAC. Patients enrolled onto this trial will be

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

response scores on the two arms using a two-tailed 0.05 significance level two group t-test. In practice, if the response scores on either disease is defined as any metastatic disease that is not extensive. High volume disease is defined as: Visceral Metastases (extranodal) and /or Bone Metastases, at least 4 or more bone lesions, one of which must be outside of the vertebral column and pelvis.) With 17 arm do not follow a normal distribution (Shapiro-Wilks test p<0.05), then the two arms will be compared by a Wilcoxon rank sum volume between the arms, patients will be stratified for low vs. high volume disease at randomization (definition: Low volume Each patient will have a response score from 0 to 30 determined (see section 1.2.5 and 6.5). To minimize differences in disease evaluable patients per arm, there would be 81% power to detect a 1.0 SD difference (effect size=1.0) between the mean of the

Another secondary objective will be to compare in the same fashion patients after completing combination or sequence therapy; thus In addition, as a secondary evaluation, patients' response scores will be compared between the two arms at 39 weeks and 1 year. PROSTVAC arm. As these comparisons will be considered exploratory, the results will be presented without correction for the response scores after 19 weeks in the docetaxel + PROSTVAC arm will be compared to 39 weeks in the docetaxel followed by comparison made at the primary time points.

applicable and the results from these analyses will be presented without formal adjustment for multiple comparisons, but in the context Antibody Response, Natural Killer (NK) Cells, Regulatory T Cells; to evaluate changes in the tumor microenvironment with biopsies pre and post (2 cycles of therapy) when feasible (biopsies could include primary tumor); and to evaluate time to progression on PET Other secondary objectives are to evaluate immunologic response including antigen-specific T-cell responses, T cell proliferation, imaging (NaF PET). These other secondary objectives will each be analyzed using appropriate nonparametric methods when of the number of such evaluations undertaken. Time to progression will be estimated using a Kaplan-Meier curve.

#### 2 ARM C

response scores on either arm do not follow a normal distribution (Shapiro-Wilks test p<0.05), then the two arms will be compared by there are 17 evaluable patients on the better of the two randomized arms, there will be 80% power to detect a 1.0 SD (effect size=1.0) Following amendment D, patients who have not been treated with 28 days of ADT will be enrolled onto a single arm (Arm C) with randomized arms. In order to do so, 26 evaluable patients without prior treatment will be enrolled onto the new arm. Assuming that a Wilcoxon rank sum test. The significance level is set at 0.025 for the second comparison since it is being added as a new primary PROSTVAC upfront followed by docetaxel. The objective for these subsequent previously untreated patients will be to obtain the comparison, and to be conservative, but the original comparison will remain at the 0.05 level since its interpretation should not be diminished by the subsequent addition of a second primary objective. Although the comparison is not based on two concurrently same 0-30 response score and to compare these scores to those obtained from the arm with superior scores from among the two difference between the means of the scores on the two arms using a 0.025 significance level two group t-test. In practice, if the

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

evaluated; if appropriate, analyses can be done to determine the similarity of traits for patients being compared with respect to factors randomized arms, the results should at least offer a suggestion of whether there is a difference or not with respect to the score that might be shown to be associated with the magnitude of the score.

As a secondary objective, the scores from the subset consisting of previously untreated patients on the superior randomized arm will be tested against the patients on the new PROSTVAC then docetaxel arm (Arm C). This comparison may be made with low power since the number of previously untreated patients on the randomized arm is expected to be limited. As this will also be a nonrandomized comparison, it will be interpreted cautiously in that context.

#### 8.3 ACCRUAL

patients in Arm C as well, the protocol ceiling will be set at 34 + 26 + 14 (allowing for up to 12 inevaluable in arms A and B together, and 2 in arm C) = 74. Based on accrual rates in the first 8 months the trial has been open, approximately 2 to 3 patients per month are Among the initial 34 randomized patients, 8 were inevaluable. Thus, additional patients will be added in amendment D in order to expected to enroll onto the trial. As a result, including the amendment, the study is expected to complete enrollment within 2 to 3 allow for the number inevaluable to date and in the future. In order to allow for the possibility of a small number of inevaluable

# COLLABORATIVE AGREEMENTS

### 1 AGREEMENT TYPE

9.1.1 Cooperative Research and Development Agreement (CRADA):

This study is conducted under a CRADA with Bavarian Nordic, Inc. (CRADA # 02377)

9.1.2 Material Transfer Agreement

A Material Transfer Agreement (Agreement # 36562-13) is in place with Epic Sciences for the studies discussed in section 5.2.2.3

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 10 HUMAN SUBJECTS PROTECTIONS

# 10.1 RATIONALE FOR SUBJECT SELECTION

assessment will be based solely on the patient's medical status. Recruitment of patients onto this study will be through standard CCR Subjects treated on this study, will be individuals with newly diagnosed metastatic castrate sensitive prostate cancer. Eligibility mechanisms. No special recruitment efforts will be conducted.

# 10.2 INCLUSION OF WOMEN AND MINORITIES

Men of all races and ethnic groups are eligible for this trial. Women are excluded as prostate cancer does not exist in this population.

## 10.3 PARTICIPATION OF CHILDREN

Men under the age of 18 will not be eligible for participation in this study based on the fact that patients under 18 are unlikely to have this disease and there are unknown toxicities in pediatric patients.

# 10.4 PARTICIPATION OF SUBJECTS UNABLE TO GIVE CONSENT

possibility, though unlikely, that subjects could become decisionally impaired. For this reason and because there is a prospect of direct impaired during the course of the study. Note: The PI or AI will contact the NIH Ability to Consent Assessment Team (ACAT) for form so that another person can make decisions about their medical care in the event that they become incapacitated or cognitively benefit from research participation (section 10.6), all subjects will be offered the opportunity to fill in their wishes for research and surrogate. For those subjects that become incapacitated and do not have pre-determined substitute decision maker, the procedures care, and assign a substitute decision maker on the "NIH Advance Directive for Health Care and Medical Research Participation" assistance in identifying and assessing an appropriate surrogate when indicated; and/or an assessment of the capacity to appoint a described in MEC Policy 87-4 and NIH HRPP SOP 14E for appointing a surrogate decision maker for adult subjects who are (a) Adults unable to give consent are excluded from enrolling in the protocol. However re-consent may be necessary and there is a evaluation as needed for the following: an independent assessment of whether an individual has the capacity to provide consent; decisionally impaired, and (b) who do not have a legal guardian or durable power of attorney, will be followed.

# 10.5 EVALUATION OF BENEFITS AND RISKS/DISCOMFORTS

Potential risks of vaccine in this patient population include the range of side effects outlined in section 11. PROSTVAC has been well tolerated in previous large trials.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 10.5.1 Alternative Approaches or Treatments

Patients will be advised verbally and in writing regarding the risks and benefits of this trial, treatment requirements, and alternative approaches to entering the trial. Written consents will be obtained.

# 10.5.2 Procedures to Eliminate or Minimize Potential Risks

as described in the monitoring schedule (Appendix A), and must have a local physician to provide long-term care and monitoring for complications. Immediate medical treatment is available at the Clinical Center, NCI, Bethesda, Maryland, for any patients who suffer physical injury as a result of participation in this study. No compensation is available, but any injury will be evaluated and treated in Scrupulous care will be taken to minimize such side effects. All patients will be given blood tests, physical examinations, and scans, This study may involve unforeseeable risks for patients, such as side effects whose exact nature and severity are unpredictable. keeping with the benefits or care to which patients are entitled under applicable regulations.

# 10.5.3 Provisions for Monitoring Data Collection to Ensure Subject Safety

As information is gathered from this trial, clinical results will be shared with patients. Laboratory and clinical data will be frequently gathered and any new significant finding(s) found during the course of the research, which may affect a patient's willingness to participate further, will be explained.

release is required by law. Records at the National Cancer Institute are maintained according to current legal requirements, and are Confidentiality of information concerning participants will be maintained, including in all publications and presentations resulting from this study. Names of participants or material identifying participants will not be released without permission, except as such made available for review, as required by the Food and Drug Administration or other authorized users, only under the guidelines established by the Federal Privacy Act.

### 10.5.4 Optional Biopsies

bleeding, infection and visceral injury) that will be explained fully during informed consent. If patients suffer any physical injury as a All care will be taken to minimize risks that may be incurred by tumor sampling. However, there are procedure-related risks (such as result of the biopsies, immediate medical treatment is available at the NCI's Clinical Center in Bethesda, Maryland. Although no compensation is available, any injury will be fully evaluated and treated in keeping with the benefits or care to which patients are entitled under applicable regulations.

## 10.5.5 Research Radiation Risks

This research study may involve exposure to radiation from a low dose CT with Sodium Fluoride PET (NaF PET) scan at baseline, annually (within 1 month) or earlier if clinically indicated (at time of PSA, clinical progression, and or radiographic progression), with

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

combined effective dose of 1.2 rem. This is below the guideline of 5.0 rem per year allowed for research subjects by the NIH Radiation Safety Committee.

## 10.6 RISKS/BENEFITS ANALYSIS

This study involves clinical research with an experimental vaccine designed to generate an immune response against antigens found in will have any clinical effect is unknown; therefore, benefit for all subjects cannot be promised from vaccine in addition to standard of prostate cancer. Patients will undergo multiple vaccinations. Side effects of the vaccine are outlined elsewhere. Whether the vaccine care (ADT+docetaxel), nor the chance of benefit accurately predicted for all patients on study. Participation in this study is voluntary, and refusal will not result in penalty or loss of benefit to which the patient is otherwise entitled.

Participation may be discontinued at any time without penalty, and the patient will be encouraged to discuss any concerns or

# 10.7 CONSENT AND ASSENT PROCESS AND DOCUMENTATION

invasive procedure will require a separate consent form. All Associate Investigators listed in this protocol who have clinical privileges benefits, and potential alternative therapies will be explained to the patient and a signed informed consent obtained. Any experimental The investigational nature and objectives of this trial, the procedures involved, and their attendant risks and discomforts, potential are permitted to obtain informed consent.

For the optional biopsy and imaging for research in the protocol, the patient will consent at the time of the procedure. If the patient refuses the optional biopsy at that time, the refusal will be documented in the medical record and in the research record.

## 10.7.1 Telephone Re-Consent Procedure

Re-consent on this study may be obtained via telephone according to the following procedure: the informed consent document will be consent. The original informed consent document will be sent back to the consenting investigator who will sign and date the consent form with the date the consent was obtained via telephone. A fully executed copy will be returned via mail for the subject's records. sent to the subject. An explanation of the study will be provided over the telephone after the subject has had the opportunity to read the consent form. The subject will sign and date the informed consent. A witness to the subject's signature will sign and date the The informed consent process will be documented on a progress note by the consenting investigator.
Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 10.7.2 Informed Consent of Non-English Speaking Subjects

is the English version of the extant IRB approved consent document. Signed copies of both the English version of the consent and the described in MAS Policy M77-2, OHSRP SOP 12, 45 CFR 46.117 (b) (2), and 21 CFR 50.27 (b) (2). The summary that will be used If there is an unexpected enrollment of a research participant for whom there is no translated extant IRB approved consent document, translated short form will be given to the subject or their legally authorized representative and the signed original will be filed in the the principal investigator and/or those authorized to obtain informed consent will use the Short Form Oral Consent Process as medical record.

Whenever possible, interpreters will be provided copies of the relevant consent documents well before the consent conversation with Unless the PI is fluent in the prospective subject's language, an interpreter will be present to facilitate the conversation. Preferably someone who is independent of the subject (i.e., not a family member) will assist in presenting information and obtaining consent. the subject (24 to 48 hours if possible). We request prospective IRB approval of the use of the short form process for non-English speaking subjects and will notify the IRB at the time of continuing review of the frequency of the use of the Short Form.

# 11 PHARMACEUTICAL INFORMATION

# 11.1 RECOMBINANT FOWLPOX-PSA(L155)TRICOMTM

Other Names: PROSTVAC-F/TRICOMTM; PROSTVAC-F

Classification: Recombinant fowlpox virus vector vaccine of the genus Avipoxvirus.

(amino acids 154-163)]. An attenuated, live, plaque-purified isolate from the POXVAC-TC strain of fowlpox virus was used as the **Product Description:** Recombinant <u>Fowlpox</u>-PSA(L155)/TRICOM<sup>TM</sup> is a recombinant fowlpox virus vector vaccine containing the 1), and LFA-3 (leukocyte function-associated antigen-3). The PSA gene coding sequence is modified to code for a single amino acid substitution [isoleucine to leucine at amino acid position 155 of the PSA antigen (designated L155)], which is designed to enhance immunogenicity. This modification occurs in a 10-mer, HLA-A2-restricted, immunodominant epitope of the antigen [designated PSA-3 stimulatory molecules is used for in vivo recombination between the plasmid vector and parental fowlpox virus genome. The genes for human PSA and three co-stimulatory molecules (designated TRICOM<sup>TM</sup>): B7.1, ICAM-1 (intercellular adhesion moleculeparental virus for this recombinant vaccine. A plasmid vector containing the modified PSA gene and the genes for the three corecombinant vaccine is manufactured by infection of primary chicken embryo dermal (CED) cells with the recombinant fowlpox

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

virus. Fowlpox virus can infect mammalian cells and express the inserted transgenes to stimulate both humoral and cellular immunity, but cannot replicate in non-avian species, making systemic infections unlikely.

## 11.1.1 How Supplied

Recombinant Fowlpox-PSA(L155)/TRICOM<sup>TM</sup> is supplied in vials containing 0.75 mL of the vaccine at a final viral concentration titer of 2 x 109 infectious units/mL formulated in phosphate-buffered saline containing 10% glycerol.

### 11.1.2 Preparation

Thaw vials completely at room temperature. Ensure the thawed contents are at the bottom of the upright vial and vortex vigorously at high power for at least ten seconds prior to dose preparation. Withdraw 0.5 mL (1 x 109 infectious units) into a 1 mL syringe for administration by subcutaneous injection.

#### 11.1.3 Storage

Store intact vials of Recombinant Fowlpox-PSA(L155)/TRICOM<sup>TM</sup> at -70°C or colder.

#### 11.1.4 Stability

Shelf-life stability studies of the intact vials are ongoing. Once the intact vials are thawed, the vaccines maintain their potency for up to 4 days when stored at 2-8°C. Do not re-freeze thawed vials. Vials of Recombinant Fowlpox-PSA(L155)/TRICOM<sup>TM</sup> are for single-use only and do not contain a preservative. Administer prepared doses as soon as possible following preparation (i.e., within one hour). If necessary, store prepared doses at 2-8°C for up to 4 hours following preparation.

## 11.1.5 Route of Administration

Recombinant Fowlpox-PSA(L155)/TRICOM<sup>TM</sup> is administered by subcutaneous injection.

## 11.1.6 Special Handling

Fowlpox virus is classified as a Biosafety Level 1 agent. These agents are not known to cause disease in healthy human adults and are of minimal potential hazard to personnel and the environment under ordinary conditions of use. Clinicians can use techniques generally acceptable for nonpathogenic material. The recombinant vaccine is a preparation of a live virus (infectious for birds) containing DNA sequences derived from the human genome. Handle the recombinant vaccine as a hazardous biological substance and

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

dispose of waste materials as hazardous biological waste, with incineration according to local institutional policy and according to local, state, and federal regulations. Healthcare workers handling the recombinant fowlpox vaccine should avoid direct contact with pet birds for at least 72 hours after working with the agent.

# Preparation, Handling and Disposal Recommendations

- .. Strictly adhere to standard microbiological practices and techniques.
- Limit/restrict access to preparation areas while dose preparation is in progress.
- Use appropriate infection control measures (e.g., thorough hand washing) after handling any materials.
- 4. Institute and follow policies for safe handling of sharps.
- Perform all dose preparations in a certified Class II biological safety cabinet, generally using procedures, guidelines and personal protective apparel used during preparation of antineoplastic agents [e.g., minimizing creation of aerosols; no eating, drinking, handling contact lenses or applying cosmetics in the work area; using appropriate personal protective apparel - gowns, sterile latex
- gloves (double-gloving is recommended), respirator masks, protective eye wear, hair cover]. Decontaminate the biological safety cabinet prior to dose preparation with sterile gauze soaked in 10% bleach solution (0.52%). sodium hypochlorite solution), or other appropriate disinfectant suitable for decontamination, rinsing, then wiping down with sterile gauze soaked in 70% alcohol. Consult specific manufacturer's recommendations with respect to disinfectant concentration, contact time and method of application. 6.
- Have all necessary supplies on-hand before beginning the preparation procedure. Develop a detailed worksheet outlining all supplies, dose calculations, and preparation procedures, and keep it available. ۲.
- Place an empty biohazard sharps container lined with a leak-proof biohazard bag in or near the biosafety cabinet to dispose of all ∞:
- 9. Transport the agent from the freezer to the work area in leak proof bag.
- should remain in contact with the surfaces for at least five minutes prior to dose preparation. Avoid exposing the virus to Wipe or spray items used for dose preparation with 70% alcohol before placing in the biological safety cabinet. Disinfectants disinfectants.
- Wipe the syringe containing the prepared dose with 70% alcohol before removing it from the biological safety cabinet; transport it in a leak proof bag or container labeled with a biohazard symbol. 11:
- Place all waste into the sharps container lined with the leak proof biohazard bag and decontaminate the biological safety cabinet again by wiping down all surfaces with sterile gauze soaked in 10% bleach solution, or other appropriate disinfectant, rinsing, then wiping down with sterile gauze soaked in 70% alcohol. Following decontamination, dispose of personal protective apparel in the biohazard safety bag. 12.
- 13. Incinerate waste according to institutional policy and according to local, state, and federal regulations.
- 14. Handle accidental spills similarly to antineoplastic spills and/or according to institutional policy.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- Prevent others from entering the area and allow aerosols time to settle (approximately 10 minutes).
- Use protective apparel, eyewear, mask, and gloves.
- Cover spills with disposable absorbent towels.
- Decontaminate the area with 10% bleach solution, or other appropriate disinfectant suitable for decontamination, allowing approximately a 20-minute contact time.
- Dispose of all waste as biohazardous waste and incinerate according to institutional policy and according to local, state, and federal regulations.
- 15. Immediately report spills and accidents resulting in overt exposure to recombinant DNA molecules to the Institutional Biosafety Committee and NIH/OSP (Office of Science Policy). Send reports to the Office of Science Policy, National Institutes of Health, 6705 Rockledge Drive, Suite 750, MSC 7985, Bethesda, MD 20892-7985. Phone (301) 496-9838; HGTprotocols@mail.nih.gov. Provide medical evaluation, surveillance, and treatment as appropriate and maintain written records of the event.

For more information about biohazard risk group classification and biohazard safety levels see:

- NIH Guidelines for Research Involving Recombinant DNA Molecules (NIH Guidelines). See current version at: http://osp.od.nih.gov/sites/default/files/NIH Guidelines.html
- Biosafety in Microbiological and Biomedical Laboratories; U. S. Department of Health and Human Services Centers for Disease Control and Prevention and National Institutes of Health. See current edition at: http://www.cdc.gov/biosafety/publications/index.htm

# Patient Care Implications and Contraindications

Cover vaccination sites with a sterile dry dressing (e.g., Telfa pad). Once the injection site is healed, no further barrier is necessary. As a precaution, protect injection sites that are exhibiting evidence of weeping, oozing or ulceration with a sterile dry dressing. In these completion with the recombinant vaccine. Instruct patients receiving fowlpox vaccines to avoid direct contact with pet birds for at circumstances, instruct patients to avoid direct contact of the injection site with susceptible individuals (e.g.; those who may be immunocompromised by disease or therapy). Instruct patients to avoid fathering a child for at least 4 months following therapy least 72 hours after vaccination or while there are any visible lesions at the injection site.

Due to the method of manufacturing (virus grown in primary chicken embryo dermal cells), patients with a history of allergy to eggs or egg products should not receive the vaccine.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

# 11.2 RECOMBINANT VACCINIA-PSA(L155)/TRICOMTM

Other Names: PROSTVAC-V/TRICOM<sup>TM</sup>; PROSTVAC-V

Classification: Recombinant vaccinia virus vector vaccine of the genus Orthopoxvirus.

stimulatory molecules is used for in vivo recombination between the plasmid vector and parental vaccinia virus genome. The virus. Vaccinia virus can infect mammalian cells and express the inserted transgenes, and is a potent immune stimulator, eliciting both a **Product Description:** Recombinant Vaccinia-PSA(L155)/TRICOM<sup>TM</sup> is a recombinant vaccinia virus vector vaccine containing the 1), and LFA-3 (leukocyte function-associated antigen-3). The PSA gene coding sequence is modified to code for a single amino acid substitution [isoleucine to leucine at amino acid position 155 of the PSA antigen (designated L155)], which is designed to enhance immunogenicity. This modification occurs in a 10-mer, HLA-A2-restricted, immunodominant epitope of the antigen [designated PSA-3 (amino acids 154-163)]. An attenuated, live, derivative of the Wyeth (New York City Board of Health) strain of vaccinia virus is used as the parental virus for the recombinant vaccine. A plasmid vector containing the modified PSA gene and the genes for the three corecombinant vaccine is manufactured by infection of primary chicken embryo dermal (CED) cells with the recombinant vaccinia strong humoral and cellular immune response. Vaccinia virus is replication competent in mammalian cells, making systemic infections genes for human PSA and three co-stimulatory molecules (designated TRICOM<sup>TM</sup>): B7.1, ICAM-1 (intercellular adhesion molecule-

## 11.2.1 How Supplied

Recombinant Vaccinia-PSA(L155)/TRICOM<sup>TM</sup> is supplied in vials containing 0.75 mL of the vaccine at a final viral concentration titer of 4 x 108 infectious units/mL formulated in phosphate-buffered saline containing 10% glycerol.

#### 11.2.2 Preparation

Thaw vials completely at room temperature. Ensure the thawed contents are at the bottom of the upright vial and vortex vigorously at high power for at least ten seconds prior to dose preparation. Withdraw 0.5 mL (2 x 108 infectious units) into a 1 mL syringe for administration by subcutaneous injection.

#### 11.2.3 Storage

Store intact vials of Recombinant Vaccinia-PSA(L155)/TRICOM<sup>TM</sup> at -70°C or colder.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

#### 11.2.4 Stability

Shelf-life studies of the intact vials are ongoing. Once the intact vials are thawed, the vaccines maintain their potency for up to 4 days when stored at 2-8°C. Do not re-freeze thawed vials. Vials of Recombinant Vaccinia-PSA(L155)/TRICOM<sup>TM</sup> are for single-use only and do not contain a preservative. Administer prepared doses as soon as possible following preparation (i.e., within one hour). If necessary, store prepared doses at 2-8°C for up to 4 hours following preparation.

## 11.2.5 Route of Administration

Recombinant Vaccinia-PSA(L155)/TRICOM<sup>TM</sup> is administered by subcutaneous injection.

## 11.2.6 Special Handling and Precautions

hazard to personnel and the environment. The recombinant vaccine is a preparation of a live virus affecting humans and contains DNA Vaccinia virus is classified as a Biosafety Level 2 agent. These agents are associated with human disease and are of moderate potential sequences derived from the human genome. Handle the recombinant vaccine as an infectious hazardous biological substance and dispose of waste materials as infectious hazardous biological waste, with incineration according to local institutional policies and according to local, state, and federal regulations.

# Preparation, Handling and Disposal Recommendations

- Prepare a biosafety manual which advises personnel of special hazards and specific instructions on practices and procedures.
- Post warning hazard signs on access doors, identifying the agents, the biosafety level, the name and phone number of the Principal Investigator or other responsible person, and any special requirements for entry.
- Establish policies and procedures allowing only personnel who are knowledgeable of the potential hazards and meet specific entry requirements (e.g., immunization) into agent preparation or storage areas.
  - Strictly adhere to standard microbiological practices and techniques.
- Limit/restrict access to preparation areas while dose preparation is in progress.
- Use appropriate infection control measures (e.g., thorough hand washing) after handling any materials.
- Institute and follow policies for safe handling of sharps. Use only needle-lock syringes and needles for dose preparation. Use extreme caution to prevent autoinoculation. Do not bend, shear, or replace the needle guard from the syringe following use. Promptly place used needles and syringes in puncture-resistant containers for disposal.

- Perform all dose preparations in a certified Class II biological safety cabinet, generally using procedures, guidelines and personal protective apparel used during preparation of antineoplastic agents [e.g., minimizing creation of aerosols; no eating, drinking, handling contact lenses or applying cosmetics in the work area; using appropriate personal protective apparel - gowns, sterile latex gloves (double-gloving is recommended), respirator masks, protective eyewear, hair cover]. ∞.
- . Perform all procedures carefully to minimize aerosol creation.
- 10. Decontaminate the biological safety cabinet prior to dose preparation with sterile gauze soaked in 10% bleach solution (0.52% sodium hypochlorite solution), or other appropriate disinfectant suitable for decontamination, rinsing, then wiping down with sterile gauze soaked in 70% alcohol. Consult specific manufacturer's recommendations with respect to disinfectant concentration, contact time and method of application.
  - 11. Have all necessary supplies on-hand before beginning the preparation procedure. Develop a detailed worksheet outlining all supplies, dose calculations, and preparation procedures, and keep it available.
    - Place an empty biohazard sharps container in the biosafety cabinet to dispose of all waste generated.
      - 3. Transport the agent from the freezer to the work area in leak proof bag.
- should remain in contact with the surfaces for at least five minutes prior to dose preparation. Avoid exposing the virus to Wipe or spray items used for dose preparation with 70% alcohol before placing in the biological safety cabinet. Disinfectants
- Wipe the syringe containing the prepared dose with 70% alcohol before removing it from the biological safety cabinet; transport it in a leak proof bag or container labeled with a biohazard symbol. 15.
- 16. Place all waste into a sharps container lined with the leak proof biohazard bag and decontaminate the biological safety cabinet again by wiping down all surfaces with sterile gauze soaked in 10% bleach solution, or other appropriate disinfectant, rinsing, then wiping down with sterile gauze soaked in 70% alcohol. Following decontamination, dispose of personal protective apparel in the biohazard safety bag.
- Place all waste and protective apparel in a leak proof biohazard bag, and place the bag inside a biohazard sharps container for incineration according to institutional policy and according to local, state, and federal regulations.
  - 18. Handle accidental spills similarly to antineoplastic spills and/or according to institutional policy:
- Prevent others from entering the area and allow aerosols time to settle (approximately 10 minutes).
  - b. Use protective apparel, eyewear, mask, and gloves.
- c. Cover spills with disposable absorbent towels.
- Decontaminate the area with 10% bleach solution, or other appropriate disinfectant suitable for decontamination, allowing approximately a 20-minute contact time.
- Dispose of all waste and protective apparel as infectious biohazardous waste and incinerate according to institutional policy and according to local, state, and federal regulations. ö

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

19. Immediately report spills and accidents resulting in overt exposure to recombinant DNA molecules to the Institutional Biosafety Committee and NIH/OSP (Office of Science Policy). Send reports to the Office of Science Policy, National Institutes of Health, 6705 Rockledge Drive, Suite 750, MSC 7985, Bethesda, MD 20892-7985. Phone (301) 496-9838; HGTprotocols@mail.nih.gov. Provide medical evaluation, surveillance, and treatment as appropriate and maintain written records of the event.

For more information about biohazard risk group classification and biohazard safety levels:

- NIH Guidelines for Research Involving Recombinant DNA Molecules (NIH Guidelines). See current version at: http://osp.od.nih.gov/sites/default/files/NIH Guidelines.html
- Biosafety in Microbiological and Biomedical Laboratories; U. S. Department of Health and Human Services Centers for Disease Control and Prevention and National Institutes of Health. See current edition at: http://www.cdc.gov/biosafety/publications/index.htm

## Precautions for Healthcare Workers

healthcare personnel from vaccine recipients have been published. If appropriate infection control precautions are observed (such as covering the vaccination site and washing hands after contact with the vaccination site or bandages), healthcare workers are probably at less risk of infection than laboratory workers because of the smaller volume and lower titers of virus in clinical specimens as participants in clinical studies must adhere to appropriate infection control measures and should be offered vaccination with the Recombinant vaccinia virus transmission risk to exposed healthcare workers is unknown. To date, no reports of transmission to compared with laboratory material. However, because of the potential risk for transmission, healthcare personnel who prepare or administer doses of recombinant vaccinia vaccine or have direct contact with contaminated dressings or other infectious material from licensed vaccinia vaccine. Do not administer routine, non-emergency vaccination with the licensed vaccinia vaccine to healthcare workers, if they, or for at least three weeks after vaccination, their close household contacts (close household contacts are those who share housing or have close physical contact):

- have active eczema or a history of eczema or atopic dermatitis, or Darier's disease.
- have other acute, chronic, or exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds), until the condition resolves.
- are pregnant or intend to become pregnant within 4 weeks of vaccination or are breast-feeding.
- are immunodeficient or immunocompromised (by disease or therapy), including HIV infection.

Additionally, do not administer routine, non-emergency vaccination with the licensed vaccinia vaccine to healthcare workers if the

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- has a moderate or severe acute illness, until the illness resolves.
- is less than 18 years of age, unless specifically indicated.
- is undergoing topical steroid therapy for inflammatory eye diseases or undergoing therapy with systemic steroids; potential immune suppression increases risk for vaccinia-related complications.
- has a history of allergy or serious reaction to prior vaccinia vaccination or any of the vaccine's components.
- cardiomyopathy, stroke or TIA) or who have  $\geq 3$  known risk factors for cardiac disease (e.g., hypertension, hypercholesterolemia, prophylactic vaccination with the licensed vaccinia vaccine while a possible causal relationship between vaccination and cardiac As a precaution, the CDC recommends that individuals with known cardiac disease (e.g., previous MI, angina, CHF, diabetes, first degree relative with onset of cardiac complications prior to age 50, smoker), not receive routine, non-emergency, events is being evaluated.

patient's inoculation site if you are pregnant or breast-feeding; have a history or presence of active eczema or atopic dermatitis; have acute, chronic or exfoliative skin conditions; or, are immunocompromised. More information on vaccinia precautions for healthcare Avoid exposure to the recombinant vaccinia vaccine, any contaminated dressings, or other infectious materials from patients, or the workers can be obtained from http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5010a1.htm#tab2 and http://www.cdc.gov/mmwr/PDF/rr/rr5207.pdf.

The CDC is the only source of the licensed vaccinia vaccine. The CDC will provide vaccinia vaccine to protect laboratory and other institution. Revaccination is recommended every 10 years. For instructions on obtaining the licensed vaccinia vaccine, contact Drug including vaccinia recombinants. The vaccine should be administered under the supervision of a physician selected by the study healthcare personnel, whose occupations place them at risk of exposure to vaccinia and other closely related orthopoxviruses, Services, National Center for Infectious Diseases, CDC at (404) 639-3670.

# Recombinant Vaccinia Vaccine Patient Care Implications, Contraindications and Potential Complications

# Patient Care Implications and Contraindications

appropriate biohazard containers. Do not administer the recombinant vaccinia vaccine if the recipient, or for at least three weeks after laundering of clothing, etc. Treat patient bandages or dressings removed from the vaccination site as infectious waste and dispose in Cover vaccination sites with a sterile dry dressing (e.g., Telfa pad). Instruct patients on proper hand-hygiene, sterile dressing care, bathing, vaccination, their close household contacts (close household contacts are those who share housing or have close physical contact):

- have active eczema or a history of eczema or atopic dermatitis, or Darier's disease.
- have other acute, chronic, or exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne, contact dermatitis, psoriasis, herpes or other open rashes or wounds), until the condition resolves.

- milk. Patients (i.e., vaccinees) should avoid fathering a child for at least 4 months following completion of therapy with the are pregnant or intend to become pregnant (due to the potential risk of fetal vaccinia); or are breast-feeding (due to the potential risk of contact transmission and inadvertent inoculation). It is currently unknown if vaccinia virus or antibodies are excreted in breast recombinant vaccine.
- are in close contact with children less than 3 years of age (due to the potential risk of contact transmission and inadvertent inoculation).
- are immunodeficient or immunocompromised (by disease or therapy), including individuals with HIV infection.

Additionally, do not administer the recombinant vaccinia vaccine if the vaccinee:

- has a moderate or severe acute illness, until the illness resolves.
- is undergoing topical steroid therapy for inflammatory eye diseases, or undergoing therapy with systemic steroids; potential immune suppression increases risk for vaccinia-related complications.
- At this time, until a more definitive causal relationship is determined, it is recommended that patients with known CHF or clinically significant cardiomyopathy, not be vaccinated with recombinant vaccinia-based vaccines, due to the potential for development of myocarditis and/or pericarditis.

Vaccination Program causes angina or heart attacks, it acknowledges a possible causal relationship between the vaccination and heart inflammation. The CDC continues to study the relationship, but in the meantime, recommends excluding individuals with underlying heart disease from participation in the current Smallpox Vaccination Program. Patients are being immunized with recombinant vaccinia vaccines with therapeutic intent and will be evaluated for cardiovascular risk factors and recent or symptomatic cardiac events per protocol eligibility criteria. Patients will be encouraged to minimize cardiovascular disease risks Although the CDC believes that there is no evidence to conclude that the licensed vaccinia vaccine used in the Smallpox and encouraged to follow risk reduction according to standard medical practice.

vaccinia vaccine to patients with a history of allergy to eggs or egg products. Do not administer the recombinant vaccinia vaccine to Due to the method of manufacturing (virus grown in primary chicken embryo dermal cells), do not administer the recombinant patients with a history of allergy or serious reaction to prior vaccinia vaccination (e.g., smallpox vaccination)

# Potential Complications Associated With Recombinant Vaccinia Vaccination

When vaccinia vaccine is administered by scarification for vaccination against smallpox, expected local reactions in individuals that have not previously been vaccinated with vaccinia include the appearance of a red papule in 3-4 days, followed by vesiculation in 5-6 days, and then the formation of a pustule on days 8-9. A large area of erythema may surround the vesicle and pustule. A crusted scab

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

usually forms by the second week and sloughs by the third week, leaving a well-formed scar. Maximal viral shedding occurs from days 4-14, but can continue until the scab is shed from the skin. Other normal local reactions can include development of local satellite lesions, regional lymphadenopathy that can persist for weeks following healing of the skin lesion, considerable local edema, and intense inflammation from the vaccination (i.e., viral cellulites), which may be confused with bacterial cellulites. Systemic symptoms typically occur between 8-10 days post-vaccination and include fever, malaise, headache, chills, nausea, myalgia, local lymphadenopathy, soreness and intense erythema surrounding the vaccination site.

central lesion that may be an ulcer or scab 6-8 days following vaccination. The response to re-vaccination depends on the degree of When administered by scarification in individuals that have previously been vaccinated with vaccinia, expected local reactions include the appearance of a clear cut pustule 6-8 days following vaccination or the development of an area of definite induration around a residual immunity following previous vaccination. Similar systemic symptoms may occur, but typically at a lower frequency.

When recombinant vaccinia vaccines are administered by intradermal, intralesional, subcutaneous or intramuscular routes of injection, milder local reactions are expected, but similar systemic symptoms may occur.

generalized vaccinia, c) eczema vaccinatum, d) progressive vaccinia (vaccinia necrosum), or e) post-vaccinial encephalitis. In a 1968 There have been a number of complications reported in the literature associated with vaccinia vaccination for smallpox. Reported ten-state survey, cases of these complications per million vaccinations in adult recipients ( $\geq 20$  years of age) of vaccinia primary complications from vaccinia vaccine when given by scarification include: a) auto-inoculation of other sites with vaccinia, b) vaccination and revaccination were:

| | Primary Vaccination | Revaccination |
|----------------------------|---------------------|---------------|
| auto-inoculation | 1.909 | 25 |
| generalized vaccinia | 212.1 | 9.1 |
| eczema vaccinatum | 30.3 | 4.5 |
| progressive vaccinia | panoda auou | 8.9 |
| postvaccinial encephalitis | pənodər ənon | 4.5 |

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Based on a 1968 national survey, the number of deaths in primary vaccinees was approximately 1 per million and the number of deaths in recipients of revaccination was approximately 0.25 per million. Deaths were most often the result of postvaccinial encephalitis or progressive vaccinia.

variables, estimated cases (number of cases per million vaccinations based on vaccination of 450,293 personnel, with a median age of adverse events in military personnel following implementation of a Smallpox Vaccination Program from the period of December 13, Information has been reported by the US Department of Defense (DoD) during the post-vaccination surveillance assessment of 2002 through May 28, 2003. Although not directly comparable to historical numbers, due to differences in multiple population 26 years and 70.5% as primary vaccinees) of these same complications per million vaccinations were:

| auto-inoculation | 107 |
|----------------------------|---------------|
| generalized vaccinia | 08 |
| eczema vaccinatum | none reported |
| progressive vaccinia | none reported |
| postvaccinial encephalitis | 2.2 |

vaccinatum, and post-vaccinial encephalitis/encephalomyelitis. The complications of vaccinia vaccination may involve a number of Generally, self-limited adverse reactions that can be serious, but not life-threatening include autoinoculation, erythematous and urticarial rashes, and generalized vaccinia. More serious life-threatening complications include progressive vaccinia, eczema

rashes usually resolve spontaneously within 2-4 days. Erythema multiforme can present as different types of lesions, including sometimes be confused with generalized vaccinia, but are generally self-limiting. Patients are usually afebrile and these benign Non-specific erythematous or urticarial rashes: These rashes can appear approximately 10 days after vaccination and may macules, papules, urticaria, and bull's eye lesions (dark papule or vesicle surrounded by a pale zone and an area of erythema). These lesions may be extremely pruritic, lasting up to four weeks. Rarely, more serious bullous erythema multiforme (Stevens-Johnson syndrome) may occur, requiring hospitalization. Vaccinia Immune Globulin (VIG) therapy is not indicated to treat

these rashes. Supportive care measures are warranted since these rashes are likely manifestations of an immune response or hypersensitivity reaction to the vaccine and are not likely to contain vaccinia virus.

- Bacterial Infection: Vaccination site infection, most likely due to staphylococcus and streptococcus normal skin flora, is rare. Onset is approximately 5 days post-vaccination and is more common in children. Appropriate antibiotic therapy is required. 7
- complications associated with vaccination and revaccination. This usually results from autoinoculation of vaccinia virus transferred from the site of the vaccination. Sites typically involved include the face, eyelids, nose, mouth, genitalia, or rectum, but can also involve the arms, legs, and trunk. Contact transmission of vaccinia, with accompanying toxicities, may occur when a recently vaccinated individual has contact with a susceptible individual. In a 1968 ten-state survey, contact transmissions were reported to occur at a rate of 27 infections per million vaccinations. The age group in which contact transmission occurred most commonly was in children \le 5 years. Eczema vaccinatum as a result of contact transmission may esult in a more severe syndrome than that seen in vaccinees, perhaps because of multiple simultaneous inoculations. About 30% of eczema vaccinatum cases reported in the 1968 ten-state survey were a result of contact transmission. It is possible that the number of cases of contact transmission would be greater in today's population, due to a largely unvaccinated patient population against smallpox. Contact transmission rarely results in postvaccinial encephalitis or progressive vaccinia. Most cases of inadvertent inoculation usually resolve without specific therapy and resolution of lesions follow the same course as the vaccination site in immunocompetent individuals. VIG can be used for severe cases involving extensive lesions or if comorbid Accidental infection is the most common complication of vaccinia vaccination, accounting for approximately 50% of all conditions exist. VIG is contraindicated in the presence of isolated keratitis due to the risk of increased corneal scarring. VIG use can be considered in cases of ocular implantation, with keratitis, if vision-threatening or if other life-threatening vaccinia-**Inadvertent Inoculation**: This can occur in the vaccinee (autoinoculation) as well as in close contacts (contact transmission). related complications exist that require VIG therapy.
- Generalized vaccinia: Generalized vaccinia (GV) is characterized by a disseminated maculopapular or vesicular rash of the vaccination site lesion. The lesions are hematogenously spread and may contain vaccinia virus. In immunocompetent for patients who are systemically ill and whose condition might be toxic or who have serious underlying immunosuppressive varying extent on any part of the body and typically develops 6-9 days after vaccination. The lesions follow the same course as individuals, the rash is generally self-limiting and requires supportive care therapy. VIG treatment can be used in severe cases 4.

were identified but only 2 reports met the case definition. More than 75% of the reports received a final diagnosis of vaccinations during 2003. Out of 38,440 vaccine recipients, 29 reports of possible GV during January 2003–December 2003 and uncommonly, early stages of progressive vaccinia or other vesicular diseases (e.g., severe chickenpox or disseminated herpes). Several publications have investigated the reporting of GV among those individuals who received smallpox The differential diagnosis of GV includes eczema vaccinatum, erythema multiforme, inadvertent inoculation at multiple sites,

vaccinia and other orthopoxviruses. Of 74 cases investigated in 753,226 smallpox vaccinations administered in December 2003 among 37,542 smallpox vaccinees. The lesions (scab and/or fluid) of seven patients were tested for vaccinia virus by use of polymerase chain reaction and/or immunohistochemistry; all were found to be negative. In addition, the postscab lesions of four of the patients were biopsied. The results from two of the biopsies suggested an allergic contact dermatitis, and results of 1ypersensitivity reaction or nonspecific rash after review by dermatologists or because laboratory results were negative for 2002 to December 2004, 50 (67.6%) met the case definition of possible GV. Cases occurred more frequently in primary vaccinees (rate, 81 per 1 million vaccinees) than in those revaccinated (rate, 32 per 1 million vaccinees). However, none met polymerase chain reaction, or skin biopsy). Twenty-one reports of postscab lesions were made between January and August one each demonstrated chronic dermatitis and squamous cell carcinoma. None of the four biopsied lesions had histologic the case definition of probable or confirmed GV, including 15 with virologically negative laboratory evaluations (e.g., culture, evidence of viropathic changes and no evidence supported smallpox vaccination as a cause for any of the lesions.

- exfoliative skin conditions. It can also occur among eczematous contacts of recently vaccinated persons. Vaccinial lesions Eczema vaccinatum: Eczema vaccinatum is a serious complication in persons with eczema and other types of chronic or generalized papular, vesicular or pustular lesions) develop on areas of the skin that are, or had at one time been, eczematous. These areas become highly inflamed and lesions may spread to healthy skin. The rash is often accompanied by fever and individuals are systemically ill. The fatality rate for untreated cases (prior to availability of VIG) has been reported from 30-40%. Following availability of VIG, mortality was reduced to approximately 7%. Early diagnosis and prompt treatment with VIG is necessary to reduce mortality. ۶.
- underlying structures. Progressive lesions may spread to other skin surfaces and to bone and viscera. Progressive vaccinia is Progressive vaccinia: Progressive vaccinia is the most serious cutaneous complication, occurring when the local vaccination associated with a high mortality rate. This complication has been seen in patients with a compromised immune system due to a congenital deficiency, lymphoproliferative disease, immunosuppressive treatment, or HIV infection. Management should lesion fails to heal and develops progressive necrosis, with destruction of large areas of skin, subcutaneous tissue, and include aggressive VIG therapy. 9
- cerebral edema, mild lymphocytic meningeal infiltration, ganglion degenerative changes and perivascular hemorrhages. Older Post-Vaccinial Encephalitis/Encephalomyelitis: Vaccinial complications affecting the CNS are unpredictable. Post-vaccinial encephalitis typically affects children < 2 years of age and is characterized by an onset of symptoms 6-10 days following vaccination, which include seizures, hemiplegia, aphasia, and transient amnesia. Histopathological changes include generalized children and adults can develop encephalitis or encephalomyelitis characterized by an onset of symptoms 11-15 days following confusion, disorientation, restlessness, delirium, drowsiness, seizures and coma. Histopathological changes include demyelination with lymphocytic infiltration, but limited cerebral edema. Mortality rates have ranged from 15-25%, with 25% vaccination, which include fever, vomiting, headache, malaise, and anorexia, progressing to loss of consciousness, amnesia, 7.

effective in treating CNS disease and is not recommended. Post-vaccinial encephalitis/encephalomyelitis are diagnoses of of patients who recover being left with varying degrees and types of neurological deficits. VIG has not been shown to be exclusion and are not believed to be a result of replicating vaccinia virus. Although no specific therapy exists, supportive care, anticonvulsants, and intensive care might be required. A review of vaccinia-related deaths (68) during a 9-year period (1959— 1966 and 1968) revealed that among first-time vaccines, 36 (52%) patients died as a result of post-vaccinial encephalitis.

- The CDC has established a National Smallpox Vaccine in Pregnancy Registry. This registry will follow women during their Fetal Vaccinia: Fetal vaccinia is a rare, but serious complication following vaccinia vaccination during pregnancy or shortly before conception (e.g., within four weeks). To date, fewer than 50 cases have been reported and often result in fetal or neonatal death. Efficacy of VIG therapy in a viable infant or used prophylactically in women during pregnancy is unknown. pregnancies and their babies, after they are born, to determine the outcome of such pregnancies. The CDC can be contacted at ∞.
- myocarditis, pericarditis, and myopericarditis. Although the CDC believes that there is no evidence to conclude that the icensed vaccinia vaccine causes angina or heart attacks, it acknowledges a possible causal relationship between the individuals with underlying heart disease be excluded from participation in the current Smallpox Vaccination Program. While t is currently not possible to fully evaluate the risk of cardiac events or the risk of myocarditis, pericarditis, or myopericarditis associated with vaccinia vaccination, it is reasonable to inform patients participating in studies using recombinant vaccinia virus of these reports and provide relevant guidance for evaluating these events. Further investigation from the ongoing Patients are being immunized with recombinant vaccinia vaccines with therapeutic intent and will be evaluated for cardiovascular risk factors and recent or symptomatic cardiac events per protocol eligibility criteria. Patients will be practice. At this time the evidence for an association with myocarditis, pericarditis, or myopericarditis seems plausible, but a rare event. If not otherwise excluded, patients with known CHF or clinically significant cardiomyopathy requiring treatment Myocarditis/Pericarditis: The CDC has recommended a temporary medical deferral to the voluntary Smallpox Vaccination Program for persons with heart disease or cardiovascular risk factors (March 25, 2003) and issued "interim supplementary information" regarding evidence that smallpox vaccination may cause myocarditis and/or pericarditis (March 31, 2003) in vaccination and heart inflammation. The CDC continues to study the relationship, but in the meantime, recommends that encouraged to minimize cardiovascular disease risks and encouraged to follow risk reduction according to standard medical people recently vaccinated with the smallpox vaccine. The cardiac events reported include myocardial infarction, angina, vaccine program may provide additional data regarding an association or lack of association with cardiovascular disease. should be excluded from protocol eligibility. 9.

Out of a total of 540,824 military personnel vaccinated with a New York City Board of Health strain of vaccinia from December 2002 through December 2003, 67 developed symptomatic myopericarditis. In the 61 ECGs that were reviewed, an identifiable abnormality was evident in 46 (75.4%). The most common abnormalities included ST-segment changes observed

follow-up of 64 patients, all patients had objective normalization of electrocardiography, echocardiography, graded exercise evident in 40 patients (65.6%); 5 patients (8.2%) had normal variant early repolarization, and T-wave abnormalities were noted in 11 patients (18.0%). In addition, cardiac enzymes were elevated in 60 of 61 (98.4%) patients evaluated with this assay. On testing, laboratory testing, and functional status; 8 (13%) reported atypical, non-limiting persistent chest discomfort. Among 37,901 health care workers vaccinated with the identical strain, 21 myo/pericarditis cases were identified; 18 (86%) were revacinees. Twelve met criteria for either myocarditis or myopericarditis, and 9 met criteria for pericarditis only (6 suspected and 3 probable). The severity of myo/pericarditis was mild, with no fatalities, although 9 patients (43%) were hospitalized

## 11.3 DOCETAXEL (TAXOTERE®)

(Please see package insert for complete drug information)

11.3.1 Source

Docetaxel will be obtained from commercial sources by the local site pharmacy.

### 11.3.2 Formulation

TAXOTERE® (docetaxel) Injection Concentrate, Intravenous infusion (IV) is a sterile, non-pyrogenic, pale yellow to brownishyellow, non-aqueous solution in single-use vials containing 20 mg docetaxel (anhydrous), 0.54 grams polysorbate 80 and 0.395 grams dehydrated alcohol solution per milliliter in two presentations:

- TAXOTERE® (docetaxel) Injection Concentrate 20 mg docetaxel in 1 mL in 50/50 (v/v) ratio polysorbate 80/dehydrated alcohol in a blister pack in one carton (NDC 0075-8003-01)
  - TAXOTERE® (docetaxel) Injection Concentrate 80 mg docetaxel in 4 mL in 50/50 (v/v) ratio polysorbate 80/dehydrated alcohol in a blister pack in one carton (NDC 0075-8004-04) 7

### 11.3.3 Preparation

Dilute the concentrated drug product:

- 1. After removing Taxotere® from refrigeration, allow them to stand at room temperature approximately 5 minutes before
- 2. Use only a 21-Gauge needle to withdraw the drug product from a vial

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

• Larger bore needles (e.g., 18 and 19 gauge) may result in stopper coring and introduce particulate matter into the drug

- Aseptically withdraw the amount of concentrated docetaxel solution required for a patient's dose with a calibrated syringe and transfer it into an appropriate parenteral product bag or bottle containing a volume of either 0.9% NS or D5W sufficient to produce a final docetaxel concentration within the range 0.3 - 0.74 mg/mL33
  - Product concentrations must not exceed 0.74 mg docetaxel per milliliter
- To minimize patient exposure to phthalate plasticizers (e.g., DEHP), which may be leached from PVC containers, prepare and store docetaxel injection for administration to patients in bottles (glass, polypropylene) or plastic bags (polypropylene,
- 4. Thoroughly mix the admixture by manual rotation and by gently inverting the product container
- When prepared as described and stored between  $2^{\circ} 25^{\circ}$ C, docetaxel solutions are stable for 4 hours

## 11.3.4 Storage and Stability

Store between 2°C and 25°C. Retain in the original package to protect from bright light. Freezing does not adversely affect the product.

## 11.3.5 Administration Procedures

To minimize patient exposure to phthalate plasticizers (e.g., DEHP), which may be leached from PVC containers and administration sets, administer docetaxel only through polyethylene-lined administration sets

## 11.3.6 Incompatibilities

- Hypersensitivity to docetaxal or polysorbate 80; neutrophil counts of <1500/μL.
- Cytochrome P450 3A4 inducers, inhibitors, or substrates: May alter docetaxel metabolism.

#### 11.3.7 Toxicity

(See package insert for complete list of side effects)

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

hypersensitivity, thrombocytopenia, neuropathy, dysgeusia, dyspnea, constipation, anorexia, nail disorders, fluid retention, asthenia, The most common adverse reactions across all docetaxel indications are infections, neutropenia, anemia, febrile neutropenia, pain, nausea, diarrhea, vomiting, mucositis, alopecia, skin reactions, myalgia.

- Siegel, R.L., K.D. Miller, and A. Jemal, Cancer statistics, 2015. CA Cancer J Clin, 2015. 65(1): p. 5-29.
- Paller, C.J. and E.S. Antonarakis, Management of biochemically recurrent prostate cancer after local therapy: evolving standards of care and new directions. Clin Adv Hematol Oncol, 2013. 11(1): p. 14-23.  $\vec{c}$
- Sweeney, C.J., et al., Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer. N Engl J Med, 2015.  $\ddot{s}$
- James, N.D., et al., Docetaxel and/or zoledronic acid for hormone-naïve prostate cancer: First overall survival results from STAMPEDE (NCT00268476). J Clin Oncol 33, 2015 (suppl; abstr 5001). 4
- Patel, P.H. and D.R. Kockler, Sipuleucel-T: a vaccine for metastatic, asymptomatic, androgen-independent prostate cancer. Ann Pharmacother, 2008. 42(1): p. 91-8. 5
- Kantoff, P.W., et al., Overall survival analysis of a phase II randomized controlled trial of a Poxviral-based PSA-targeted immunotherapy in metastatic castration-resistant prostate cancer. J Clin Oncol, 2010. 28(7): p. 1099-105. 6.
- Longo, D.L., New therapies for castration-resistant prostate cancer. N Engl J Med, 2010. 363(5): p. 479-81. 7.
- Madan, R.A., et al., Prostvac-VF: a vector-based vaccine targeting PSA in prostate cancer. Expert Opin Investig Drugs, 2009. **18**(7): p. 1001-11.  $\infty$
- Arlen, P.M., et al., Clinical safety of a viral vector based prostate cancer vaccine strategy. J Urol, 2007. 178(4 Pt 1): p. 1515-9.
- Gulley, J.L., et al., Immunologic and prognostic factors associated with overall survival employing a poxviral-based PSA vaccine in metastatic castrate-resistant prostate cancer. Cancer Immunol Immunother, 2010. 59(5): p. 663-74. 10.
- Garnett, C.T., J. Schlom, and J.W. Hodge, Combination of docetaxel and recombinant vaccine enhances T-cell responses and antitumor activity: effects of docetaxel on immune enhancement. Clin Cancer Res, 2008. 14(11): p. 3536-44. 11.
- Hodge, J.W., et al., Chemotherapy-induced immunogenic modulation of tumor cells enhances killing by cytotoxic T ymphocytes and is distinct from immunogenic cell death. Int J Cancer, 2013. 133(3): p. 624-36. 12.
- Madan, R.A., P.M. Arlen, and J.L. Gulley, PANVAC-VF: poxviral-based vaccine therapy targeting CEA and MUC1 in carcinoma. Expert Opin Biol Ther, 2007. 7(4): p. 543-54. 13.
- Heery, C.R., et al., A Phase 2 Randomized Trial of Docetaxel Alone or in Combination with a Therapeutic Cancer Vaccine PANVAC) in Patients with Metastatic Breast Cancer JAMA Oncology, in press 14.

- Stein, W.D., et al., Tumor growth rates derived from data for patients in a clinical trial correlate strongly with patient survival: a novel strategy for evaluation of clinical trial data. Oncologist, 2008. 13(10): p. 1046-54. 15.
- Stein, W.D., et al., Bevacizumab reduces the growth rate constants of renal carcinomas: a novel algorithm suggests early discontinuation of bevacizumab resulted in a lack of survival advantage. Oncologist, 2008. 13(10): p. 1055-62. 16.
- Stein, W.D., et al., Tumor regression and growth rates determined in five intramural NCI prostate cancer trials: the growth rate constant as an indicator of therapeutic efficacy. Clin Cancer Res, 2011. 17(4): p. 907-17. 17.
- Madan, R.A., et al., Clinical evaluation of TRICOM vector therapeutic cancer vaccines. Semin Oncol, 2012. 39(3): p. 296-18.
- Hodi, F.S., et al., Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med, 2010. 363(8): p. 19.
- Madan, R.A. and J.L. Gulley, (R)Evolutionary therapy: the potential of immunotherapy to fulfill the promise of personalized cancer treatment. J Natl Cancer Inst, 2015. 107(1): p. 347. 20.
- Chen, D.S. and I. Mellman, Oncology meets immunology: the cancer-immunity cycle. Immunity, 2013. 39(1): p. 1-10. 21.
- Disis, M.L., et al., Concurrent trastuzumab and HER2/neu-specific vaccination in patients with metastatic breast cancer. J Clin Oncol, 2009. 27(28): p. 4685-92. 22.
- Walter, S., et al., Multipeptide immune response to cancer vaccine IMA901 after single-dose cyclophosphamide associates with longer patient survival. Nat Med, 2012. 18(8): p. 1254-61. 23.
- Hardwick, N. and B. Chain, Epitope spreading contributes to effective immunotherapy in metastatic melanoma patients. Immunotherapy, 2011. **3**(6): p. 731-3. 24.
- Iu, S., et al., CD13+CD4+CD25hi regulatory T cells exhibit higher suppressive function and increase with tumor stage in non-small cell lung cancer patients. Cell Cycle, 2009. 8(16): p. 2578-85. 25.
- Vergati, M., et al., Analysis of circulating regulatory T cells in patients with metastatic prostate cancer pre-versus postvaccination. Cancer Immunol Immunother, 2011. **60**(2): p. 197-206. 26.
- Sharifi, N., et al., A polymorphism in a transporter of testosterone is a determinant of androgen independence in prostate cancer. BJU Int, 2008. 102(5): p. 617-21. 27.
- Hamada, A., et al., Effect of SLCO1B3 haplotype on testosterone transport and clinical outcome in caucasian patients with androgen-independent prostatic cancer. Clin Cancer Res, 2008. 14(11): p. 3312-8. 28.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

- scintigraphy, single- and multi-field-of-view SPECT, 18F-fluoride PET, and 18F-fluoride PET/CT. J Nucl Med, 2006. 47(2): p. Even-Sapir, E., et al., The detection of bone metastases in patients with high-risk prostate cancer: 99mTc-MDP Planar bone 29.
- Even-Sapir, E., et al., 18F-Fluoride positron emission tomography and positron emission tomography/computed tomography Semin Nucl Med, 2007. 37(6): p. 462-9. 30.
- Eisenhauer, E.A., et al., New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer, 2009. 45(2): p. 228-47. 31.
- testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol, 2008. 26(7): p. 1148-59. Scher, H.I., et al., Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of 32.
- Bubley, G.J., et al., Eligibility and response guidelines for phase II clinical trials in androgen-independent prostate cancer: recommendations from the Prostate-Specific Antigen Working Group. J Clin Oncol, 1999. 17(11): p. 3461-7. 33.
- Rustin, G.J., et al., Re: New guidelines to evaluate the response to treatment in solid tumors (ovarian cancer). J Natl Cancer Inst, 2004. 96(6): p. 487-8. 34.
- Vergote, I., et al., Re: new guidelines to evaluate the response to treatment in solid tumors [ovarian cancer]. Gynecologic Cancer Intergroup. J Natl Cancer Inst, 2000. 92(18): p. 1534-5. 35.

## 13 APPENDIX A: STUDY CALENDAR

# ARM A: Sequential Docetaxel followed by PROSTVAC

| | Screening/ | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | W | Safety | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline <sup>7</sup> | -7 | 1 | 4 | 7 | | 13 | 16 | 19 | 21 | 24 | 27 | 30 | | Ą | Visit | q 12 weeks |
| | | | | | | | | | | | | | | | 36 | | until |
| | | | | | | | | | | | | | | | | | disease |
| | | | | | | | | | | | | | | | | | progression |
| Treatment | | | | | | | | | | | | | | | | | |
| Vaccinia- | | | | | | | | | X | | | | | | | | |
| PROSTVAC | | | | | | | | | | | | | | | | | |
| Fowlpox- | | | | | | | | | | X | X | X | X | X | X | | |
| PROSTVAC | | | | | | | | | | | | | | | | | |
| Docetaxel (75 | | | X | X | X | X | X | X | | | | | | | | | |
| $ mg/m^2)^1$ | | | | | | | | | | | | | | | | | |


| Follow-up<br>q 12 weeks<br>until<br>disease<br>progression | X | | X | | | | | X | | $X^9$ | | | $X_8$ | $X_8$ | X | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety<br>Visit | | | X | | | | | × | | X | | | | | | X | X |
| W k | | | X | | | | | × | | | | | | | | X | X |
| Wk<br>33 | 50 | | X | | | | | × | | | | | | | | X | X |
| Wk<br>30 | dosing | | X | | | | | × | | | | | | | | X | × |
| Wk 27 | revious | | X | | | | | X | | | | | | | | X | X |
| Wk 24 | Continued at standard schedule based on patients previous dosing | | X | | | | | × | | X | X | | | | | X | × |
| Wk 21 | d on pa | | X | | | | | × | | | | | | | | X | X |
| Wk<br>19 | le base | | X | | | | | × | | X | | | × | × | | X | X |
| Wk<br>16 | schedu | | X | | | | | × | | | | | | | | X | × |
| Wk<br>13 | andard | | X | | | | | × | | X | | | | | | X | × |
| Wk<br>10 | ed at st | | X | | | | | × | | X | | | | | | X | × |
| Wk<br>7 | Continu | | X | | | | | × | | | | | | | | X | X |
| Wk<br>4 | ) | | X | | | | | X | | | | | | | | X | X |
| Wk<br>1 | | | X | | | | | X | | X | | X | | | | X | X |
| Wk2 | | | | | | | | | | | | | | | | X | × |
| Screening/<br>Baseline <sup>7</sup> | | | $X^{3,4}$ | $X^{3,4}$ | | $X^2$ | | X <sup>3,4</sup> | | X | X | | X <sub>3</sub> | X <sub>3</sub> | × | | |
| | GnRH Agonist/<br>Antagonist | Assessments | History and PE,<br>Ht and Wt | ECOG | Performance<br>Score and ECG | Pathologic | confirmation of dx <sup>2</sup> | Labs (see section | <b>2.2</b> and <b>2.3</b> ) | Research Bloods | Biopsy (optional) | PΚ <sup>5</sup> | Tc 99<br>scintigraphy | CT-C/A/P, or<br>MRI | Experimental Imaging (optional) <sup>6</sup> | Adverse Events | Concomitant<br>Medications |

<sup>1</sup>Docetaxel will be given with dexamethasone premedication: Dexamethasone 8 mg PO for 3 doses at 12 h, 3 h, & 1 h before starting docetaxel

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

 $\overline{\text{OR}}$  Dexamethasone 12 mg IV 30 – 60 min before docetaxel for patients who miss  $\geq 1$  oral dexamethasone doses

<sup>2</sup>Pathologic confirmation will be obtained any time prior to initiation of study therapy

<sup>3</sup>Screening assessments obtained within 8 weeks prior to initiation of study therapy

'Baseline assessments obtained within 16 days prior to initiation of study therapy (these tests will not need to be repeated if they were done at screening within the appropriate timeframe)

<sup>5</sup>Required unless logistically not feasible:

Blood samples for the determination of docetaxel (DTX) plasma levels will be obtained from participating patients via 6mL sodium heparin tube (BD, Franklin Lakes, NJ) collected just prior to drug administration (predose), 5-min prior to end of 1-hr infusion (or just prior to infusion end), then 15min, 30min, 3hr, 6hr, 12hr, and 24hr post end of infusion (EOI). Blood draws will be permitted to have a window of +/- 5min to accommodate logistical challenges. Samples will be obtained from patients only during first dose of DTX on both study arms. Bioanalytical measurements will be conducted on an ultra HPLC-MSMS system by the Clinical Pharmacology Program (CPP).

This data will be used to monitor DTX plasma accumulation for pharmacokinetic analysis and in order to assess any drug-vaccine interactions or correlations, as well as correlations with pharmacogenomics, adverse events, and clinical response.

When logistically feasible and with the patient's consent, experimental imaging including NaF PET, will be done at baseline, annually (within 1 month) or earlier if clinically indicated (at time of PSA, clinical progression, and or radiographic progression)

See sections 2.2 and 2.3 for screening and baseline procedures respectively

<sup>3</sup>CT and Bone scan yearly (+/- 6 weeks) from end of chemo and at serological progression as defined in Section 6.3

# **ARM B: Combined Docetaxel with PROSTVAC**

| | Screening/ Week -2 Baseline <sup>7</sup> | Week -2 | Week 1 | Week 4 | Week 7 | Week 10 | Week 13 | Week 1 Week 4 Week 7 Week 10 Week 13 Week 16 Safety Visit | Safety<br>Visit | Follow-up<br>q 12 weeks<br>until<br>disease<br>progression |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | | | | | | | | | | |
| Vaccinia- | | X | | | | | | | | |
| PROSTVAC | | | | | | | | | | |
| Fowlpox- | | | X, D1 | | X, D1 X, D1 | X, D1 | X, D1 X, D1 | X, D1 | | |
| PROSTVAC | | | | | | | | | | |
| Docetaxel (75 | | | X | X | X | X | X | X | | |
| $mg/m^2)^1$ | | | D2 or D3 | D2 or D3 | D2 or D3 | D2 or D3 D2 or D3 D2 or D3 D2 or D3 D2 or D3 D2 or D3 | D2 or D3 | D2 or D3 | | |
| GnRH | | | Contin | ued at standa | ard schedule | Continued at standard schedule based on patients previous dosing | ients previous | s dosing | | × |

<sup>&</sup>lt;sup>9</sup>Every 6 months after completion of therapy.


| | | | | | | | | | | | | , | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Follow-up q 12 weeks until disease progression | | | X | | | | | | X | | $X^9$ | | | $X_8$ | $X^8$ | X | | X | X |
| Safety<br>Visit | | | X | | | | | | X | | X | | | X | X | | | X | X |
| Week 16 | | | X | | | | | | X | | | | | | | | | X | X |
| Week 13 | | | X | | | | | | X | | X | | | | | | | X | X |
| Week 10 | | | X | | | | | | X | | | | | | | | | X | X |
| Week 7 | | | X | | | | | | X | | | | | | | | | X | X |
| Week 4 | | | X | | | | | | X | | X | X | | | | | | X | X |
| Week 1 | | | X | | | | | | X | | X | | X | | | | | X | X |
| Week -2 | | | | | | | | | | | | | | | | | | X | X |
| Screening/<br>Baseline <sup>7</sup> | | | $X^{3,4}$ | | $X^{3,4}$ | | ZX | | $X^{3,4}$ | | X | X | | ${}_{arepsilon X}$ | ${}_{arepsilon X}$ | X | | | |
| | Agonist/Antagonist | Assessments | History and PE, | Height and Weight | ECOG Performance | Score and ECG | Pathologic | confirmation of dx <sup>2</sup> | Labs (see section | <b>2.2</b> and <b>2.3</b> ) | Research Bloods | Biopsy (optional) | PK studies <sup>5</sup> | Tc 99 scintigraphy | CT-C/A/P, or MRI | Experimental | Imaging (optional) <sup>6</sup> | Adverse Events | Concomitant<br>Medications |

for 3 doses at 12 h, 3 h, & 1 h before starting docetaxel OR Dexamethasone 12 mg IV 30 – 60 min before docetaxel for patients who miss  $\geq 1$  oral Docetaxel will be given 20-48 hours after vaccine dose. Docetaxel will be given with dexamethasone premedication: Dexamethasone 8 mg PO dexamethasone doses

<sup>&</sup>lt;sup>2</sup>Pathologic confirmation will be obtained any time prior to enrollment

<sup>&</sup>lt;sup>3</sup>Screening assessments obtained within 8 weeks prior to enrollment

<sup>&</sup>lt;sup>4</sup>Baseline assessments obtained within 16 days prior to enrollment (these tests will not need to be repeated if they were done at screening within the appropriate timeframe)

<sup>&</sup>lt;sup>5</sup>Required unless logistically not feasible:

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

heparin tube (BD, Franklin Lakes, NJ) collected just prior to drug administration (predose), 5-min prior to end of 1-hr infusion (or just prior to infusion end), then 15min, 30min, 3hr, 6hr, 12hr, and 24hr post end of infusion (EOI). Blood draws will be permitted to have a window of +/-Blood samples for the determination of docetaxel (DTX) plasma levels will be obtained from participating patients via 6mL sodium 5min to accommodate logistical challenges. Samples will be obtained from patients only during first dose of DTX on both study arms. Bioanalytical measurements will be conducted on an ultra HPLC-MSMS system by the Clinical Pharmacology Program (CPP)

This data will be used to monitor DTX plasma accumulation for pharmacokinetic analysis and in order to assess any drug-vaccine interactions or correlations, as well as correlations with pharmacogenomics, adverse events, and clinical response. When logistically feasible and with the patient's consent, experimental imaging including NaF PET, will be done at baseline, annually (within 1 month) or earlier if clinically indicated (at time of PSA, clinical progression, and or radiographic progression)

See sections 2.2 and 2.3 for screening and baseline procedures respectively

CT and Bone scan yearly (+/- 6 weeks) from end of chemo and at serological progression as defined in Section 6.3

<sup>9</sup>Every 6 months after completion of therapy.


ARM C: PROSTVAC prior to Docetaxel

| p se | | | | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Follow-up<br>q 12 weeks<br>until disease<br>progression | | | | | | | | | X | | | | | × | | $X^9$ | | | $_{L}X$ | $\mathbf{X}^{7}$ | X | | | X | | × |
| Safety<br>Visit | | | | | | pa | | | X | | | | | × | | X | | | X | X | | | | X | | X |
| Chemo Wk 16 | | | | | X | as initiat | | | X | | | | | × | | | | | | | | | | X | | X |
| Chemo Wk 13 | | | | | X | ADT wa | | | × | | | | | × | | | | | | | | | | X | | X |
| Chemo WK 10 | | | | | X | when / | | | X | | | | | × | | X | | | | | | | | X | | X |
| Chemo WK | | | | | X | en and | | | X | | | | | × | | | | | | | | | | X | | × |
| Chemo Wk 4 | | | | | X | ity chos | <b>.</b> | | X | | | | | × | | | | | | | | | | X | | X |
| Chemo Wk | | | | | X | modal | | | X | | | | | × | | X | | X | $X^8$ | $X_8$ | | | | X | | X |
| Vaccine WK 15 PI discretio | | | | × | | ased on | | | X | | | | | × | | | X | | | | | | | | | X |
| Vaccine WK 12 PI discretio | | | | × | | Continued at standard schedule based on modality chosen and when ADT was initiated | | | × | | | | | × | | | | | | | | | | X | | × |
| Vaccine WK | | | | × | | ndard sc | | | X | | | | | × | | X | | | | | | | | X | | X |
| Vaccine WK | | | | × | | ed at sta | | | X | | | | | × | | X | | | | | | | | X | | X |
| Vaccine WK | | | | × | | Continu | | | X | | | | | × | | | | | | | | | | X | | X |
| Vaccine WK | | X | | | | | | | | | | | | | | | | | | | | | | X | | X |
| Screening/<br>Baseline <sup>6</sup> | | | | | | | | | $X^{2,3}$ | | $X^{2,3}$ | X | | $X^{2,3}$ | | X | X | | $X^2$ | $X^2$ | X | | | | | |
| | Treatment | Vaccinia- | PROSTVAC | Fowlpox-<br>PROSTVAC | Docetaxel (75 mg/m <sup>2</sup> ) | GnRH | Agonist/Antagonist | Assessments | History and PE, | Height and Weight | ECOG and ECG | Pathologic | confirmation of dx | Labs (see section | 2.2 and 2.3) | Research Bloods | Biopsy (optional) | PK studies <sup>4</sup> | Tc 99 scintigraphy | CT-C/A/P, or MRI | Experimental | Imaging | (optional) <sup>5</sup> | Concomitant | Medications | Adverse Events |

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

Pathologic confirmation will be obtained any time prior to enrollment

<sup>2</sup>Screening assessments obtained within 8 weeks prior to enrollment

<sup>3</sup>Baseline assessments obtained within 16 days prior to enrollment (these tests will not need to be repeated if they were done at screening within the appropriate timeframe)

<sup>4</sup>Required unless logistically not feasible:

infusion end), then 15min, 30min, 3hr, 6hr, 12hr, and 24hr post end of infusion (EOI). Blood draws will be permitted to have a window of +/-5 heparin tube (BD, Franklin Lakes, NJ) collected just prior to drug administration (predose), 5-min prior to end of 1-hr infusion (or just prior to Blood samples for the determination of docetaxel (DTX) plasma levels will be obtained from participating patients via 6mL sodium minutes to accommodate logistical challenges. Samples will be obtained from patients only during first dose of DTX on allstudy arms. Bioanalytical measurements will be conducted on an ultra HPLC-MSMS system by the Clinical Pharmacology Program (CPP)

This data will be used to monitor DTX plasma accumulation for pharmacokinetic analysis and in order to assess any drug-vaccine interactions or correlations, as well as correlations with pharmacogenomics, adverse events, and clinical response. <sup>5</sup>When logistically feasible and with the patient's consent, experimental imaging including NaF PET, will be done at baseline, annually (within 1 month) or earlier if clinically indicated (at time of PSA, clinical progression, and or radiographic progression)

<sup>6</sup>See sections 2.2 and 2.3 for screening and baseline procedures respectively

CT and Bone scan yearly (+/- 6 weeks) from end of chemo and at serological progression as defined in Section 6.3

May be performed any time within 3 weeks of first doxectaxel dose, regardless of last vaccine.

Every 6 months after completion of therapy.

#### 14 APPENDIX B: PERFORMANCE STATUS CRITERIA

| ECC | OG Performance Status Scale | Kai | rnofsky Performance Scale |
|---|---|---|---|
| Grade | Descriptions | Percent | Description |
| | Normal activity. Fully active, | 100 | Normal, no complaints, no evidence of disease. |
| 0 | able to carry on all pre-disease performance without restriction. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able | 80 | Normal activity with effort; some signs or symptoms of disease. |
| 1 | to carry out work of a light or sedentary nature (e.g., light housework, office work). | 70 | Cares for self, unable to carry on normal activity or to do active work. |
| 2 | In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out | 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| | any work activities. Up and about more than 50% of waking hours. | 50 | Requires considerable assistance and frequent medical care. |
| | In bed >50% of the time. | >50% of the time. 40 Disabled, required and assistance. | |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. | 30 | Severely disabled, hospitalization indicated. Death not imminent. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any | 20 | Very sick, hospitalization indicated. Death not imminent. |
| 4 | self-care. Totally confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. |
| 5 | Dead. | 0 | Dead. |

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

#### 15 APPENDIX C: VACCINIA-PROSTVAC PATIENT INSTRUCTION SHEET

1. What vaccination site reactions can you expect?

- 2. How should you care for the vaccination site?
- 3. Are there any activities I should avoid?
- 4. What about contact with other people?
- 5. Who do I contact when I have a question?

#### 1. What vaccination site reactions can you expect?

A typical reaction in a patient who has been previously vaccinated with vaccinia includes the appearance of a small swelling in 2-3 days that may enlarge to 1-2 inches across, a small blister or pustule after 5-7 days, and healing with little scarring within 2-3 weeks. Some patients may have very little skin reaction. Often the leg that received the vaccine may become swollen. Swollen or tender lymph nodes ("glands") in the groin may be felt. A fever to 100-101°F may occur on the second or third day. You may notice that you feel tired for 3 or 4 days. The vaccination site may itch for about 2 weeks while the scab is forming. You can take acetaminophen ("Tylenol") if you have any aches or fever but you should avoid aspirin. If fever continues for more than a day or two, you should call to speak to the clinic nurse or the research nurse.

In patients who have never received vaccinia or in some who received it a very long time ago, a red swelling is followed by a blister on day 5 to 6 and then the formation of a pustule (or "boil") 1-2 inches in diameter on day 9 to 11. A large area of redness may surround this area. A crusted scab usually forms by the second week and falls off by the third week leaving a scar roughly 1/2 inch in diameter. Fever and malaise (the "blahs") may occur during the blister and pustular phases. Swollen and tender lymph nodes may persist for months. Many of the local toxicities described (e.g., pustule and scab formation) are typical of reactions seen when vaccinia is administered via scarification or intradermal administration. These reactions may be seen, but are usually not seen when administered via subcutaneous injection.

#### 2. How should you care for the vaccination site?

Live vaccinia virus is in skin cells at the vaccination site during the 1-2 weeks until healing has occurred. Maximal viral "shedding" from the vaccination site occurs from days 4-14, but can continue until the scab falls off from the skin. After that there is no vaccinia virus in your body. You can spread the virus to other parts of your body or to other people by touching the vaccination site and then touching your eyes, mouth, a cut or some other break in the skin. You do not pass vaccinia virus by coughing or sneezing or by sharing food or cups and dishes.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

In general, frequent careful hand washing by you and by any persons in physical contact with you is the best way to prevent transmission of virus. You should also use two types of barriers over your vaccination site at all times until the scab is gone. These barriers are (1) the bandage and (2) clothing (pants or elbow length sleeves depending on the site of vaccination). These barriers should remain in place until the scab has fallen off.

For dressing care you will have a bag with some no-stick "First-Aid" or "Telfa" pads, disposable gloves, and zip-lock plastic bags. If you run out of supplies between visits, you can use a dry sterile bandage (gauze or "First-Aid" or "Telfa") from the drug store.

The no-stick pad ("First-Aid" or "Telfa" pad) dressing should be worn until the site has healed. If it remains clean and dry and is not coming off, you do not need to change it. If the dressing gets wet either from drainage from the vaccination or from water when you are showering or if it starts coming off, you should remove it and put on a clean bandage. Wear the gloves when handling the old dressings. Put the old dressing and the gloves in the zip-lock bag, then wash your hands, put on the new bandage, and wash your hands again. You do not need to wear gloves for the new bandage. You do not need to wash the vaccination site, but while the dressing is off, you may wash it lightly with a cloth, soap, and water. If you do wash, blot the site dry with a towel (don't rub), then put the wash cloth and the towel in the laundry. Do not let the shower run on the non-bandaged site because live virus could be washed onto other areas of your body. Do not put any steroid cream, medicated creams, or other ointments on the vaccination site.

Before you throw away the zip-lock bag with the old dressing and gloves in it, pour a little bleach (about a quarter cup) in the bag to help kill any virus.

Wash your hands after each step.

#### 3. Are there any activities I should avoid or take special care?

You should not go swimming until the vaccination site has healed and you no longer need to wear a bandage on it.

If you wear contact lenses, have removable dentures, have a colostomy or any other "open" area on your body that needs daily care, always wash your hands very well before handling your contact lenses, dentures, dressings, etc. Take care of all of these procedures before changing your vaccination dressing.

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

#### 4. What about contact with other people?

Remember, frequent careful hand washing by you and by any persons with whom you have physical contact is the best way to prevent transmission of virus. During the time you need to wear a bandage (for a minimum of 3 weeks after vaccination) there are several kinds of people with whom you should avoid close contact. "Close contact" means that you sleep in the same bed with the person, give the person baths, and/or touch their bare skin to change their clothes (or diapers), apply ointments, or change their bandages.

The individuals you should avoid include children ≤ 3 years of age; pregnant women or nursing women; individuals with eczema, history of eczema or other skin conditions such as active cases of extensive psoriasis, severe rashes, generalized itching, infections, burns, chicken pox, or skin trauma; and/or immune suppressed individuals such as individuals with leukemia or lymphoma, with AIDS, or those receiving immunosuppressive treatment (for example, after organ transplant).

#### 5. Who do I contact when I have a question?

If you have any questions at any time, please call. A nurse or a physician is available 24 hours a day by telephone. To speak with the research nurse, call the research nurse's office during regular business hours; if your question is not urgent, you may leave a message for the research nurse on the answering machine. If your question is urgent or if you have a question outside of the regular business hour, please contact the 3NW inpatient unit and speak with the charge nurse.

In an emergency, call 911 or report to the local emergency room/urgent care center. If you have to go to an emergency room, please ask the doctors to call NIH for more information.

#### PHONE NUMBERS

| 3NW Inpatient unit | (301) 451-0789 |
|----------------------------|------------------|
| 12th floor Oncology Clinic | (301) 496-4026 |
| Ravi Madan, MD | (301) 480-7168 * |
| James Gulley, MD, PhD | (301) 480-7164 * |

<sup>\*</sup>after regular business hours, please contact 3NW inpatient unit.

#### 16 APPENDIX D: GUIDELINES FOR PROPHYLAXIS AND TREATMENT FOR HYPERSENSITIVITY REACTIONS (HSR) ASSOCIATED WITH DOCETAXEL

| Initial Regimen | HSR Interventions Step 1 | HSR Interventions Step 2 | HSR Interventions Step 3 |
|---|---|---|---|
| For ALL patients who have not experienced an HSR associated with Docetaxel | For pts with a<br>H/O a single<br>HSR episode | For pts who experience<br>a HSR after<br>implementing Step 1<br>interventions | For pts with severe or repeated HSR episodes after implementing Steps 1 & 2 interventions |
| PREMEDICATION WITH: <b>Dexamethasone</b> 8 mg PO for 3 doses at 12 h, 3 h, & 1 h before starting docetaxel OR <b>Dexamethasone</b> 12 mg IV 30 − 60 min before docetaxel for patients who miss ≥1 oral dexamethasone doses • Reference: study protocol, Section 3.2.3 | & 3 h before starting + Dexamethasone 12 starting docetaxel + Diphenhydramine 30 min before startin + | mg PO for 2 doses at 12 h g docetaxel mg IV 30 – 60 min before 50 mg IV push 15 – | PREMEDICATION WITH: Dexamethasone 8 - 20 mg PO for 2 doses between 24 - 36 h and at 12 hours before starting docetaxel + Dexamethasone 20 mg IV 30 - 60 min before starting docetaxel + Diphenhydramine 50 - 150 mg IV push 15 - 30 min before starting docetaxel + Ranitidine 50 mg IV infusion 15 - 30 min before starting docetaxel |
| <b>Docetaxel</b> 75 mg/m <sup>2</sup> * IV over 60 minutes† | <b>Docetaxel</b> 75 mg/m <sup>2</sup> * IV over 1 – 2 hours† | Docetaxel 75 mg/m <sup>2</sup> * IV over 4 hours • Given in two portions‡, as: Docetaxel 37.5 mg/m <sup>2</sup> IV over 2 hours, q.2 h for 2 doses | <ul> <li>Docetaxel 75 mg/m²* IV</li> <li>Given in three portions‡, as follows:</li> <li>Docetaxel 5 mg in 10 mL IV via syringe pump over 60 min, followed immediately afterward by:</li> <li>Docetaxel 25 mg in 50 mL IV over 60 min, followed immediately afterward by:</li> <li>Docetaxel 75 mg/m² (minus 30 mg) IV over 120 min</li> </ul> |

#### **PRN Orders:**

Hydrocortisone 100 mg IV push q.15 min for 2 doses, PRN docetaxel reaction

+

Abbreviated Title: Docetaxel & PROSTVAC in mCSPC

| Initial Regimen | HSR Interventions Step 1 | HSR Interventions Step 2 | HSR Interventions Step 3 |
|---|---|---|---|
| For ALL patients who have not experienced an HSR associated with Docetaxel | _ | For pts who experience<br>a HSR after<br>implementing Step 1<br>interventions | = |

Diphenhydramine 50 mg IV push q.15 min for 2 doses, PRN docetaxel reaction

+

Ranitidine 50 mg IV, PRN docetaxel reaction

H

Hydromorphone 1 mg IV push q.15 min for 4 doses, PRN pain with docetaxel reaction

+

Aluminum Hydroxide 200 mg + Magnesium Hydroxide 200 mg + Simethicone 20 mg chewable tablet

1 – 2 tablets q.3 hours, PRN epigastric discomfort (drug name in CRIS is cross-referenced with "Mylanta")

† For each docetaxel product, drug delivery will be attempted over the administration period indicated, but rate titration is permitted. If rate titration is needed to accommodate patient tolerance, the following escalation scheme is recommended:

| Initial Rate: | 25 mL/h for 5 minutes |
|-----------------|--------------------------|
| Rate Escalati | on Steps: |
| 1 <sup>st</sup> | 50 mL/h for 5 minutes |
| 2 <sup>nd</sup> | 100 mL/h for 5 minutes |
| 3 <sup>rd</sup> | 200 mL/h for 5 minutes |
| 4 <sup>th</sup> | 250 mL/h until completed |

‡ Docetaxel stability is concentration dependent. All docetaxel products diluted within the range 0.3 – 0.74 mg/mL are labeled to expire 4 hours after preparation was completed.

<sup>\*</sup> Initial (unmodified) docetaxel dosage is identified. Consult the study protocol or a medically responsible investigator to determine whether docetaxel dose/dosage modification is indicated.